# Protocol LOXO-BTK-21050 (J2N-OX-JZNV) Version 1.0

A Phase I, Open-Label, Randomized, 2-Way Crossover Study to Compare the PK of Pirtobrutinib (LOXO-305) Tablets

NCT06258174

Approval date: 31-Aug-2021

# **Protocol**

# A Phase I, Open-Label, Randomized, 2-Way Crossover Study to Compare the PK of Pirtobrutinib (LOXO-305) Tablets

Protocol Status: Final Protocol Version: 1.0 Protocol Date: 31 August 2021

Investigational Medicinal Product: Pirtobrutinib

Protocol Reference: LOXO-BTK-21050 Labcorp Drug Development Study: 8478595 IND Number: 139876

Sponsor:

Loxo Oncology, Inc.

A wholly owned subsidiary of Eli Lilly and

Company

701 Gateway Boulevard, Suite 420 South San Francisco, CA 94080

USA

Coordinating Investigator Study Site: Labcorp Clinical Research Unit Inc.

3402 Kinsman Boulevard Madison, WI 53704

**USA** 

Up to 2 additional sites in the United States

may be utilized.

Sponsor Signatory:

PPD MD, PhD

Coordinating Investigator:

PPD MD

Information described herein is confidential and may be disclosed only with the express written permission of the Sponsor.

# **SPONSOR APPROVAL**

I have read the protocol and approve it:



01-Sep-21 | 14:37:26 EDT

Date

PPD MD, PhD

Medical Manitor Consultin

Medical Monitor, Consulting to Loxo Oncology, Inc.

Protocol

Labcorp Drug Development Study: 8478595

CONFIDENTIAL

Protocol Reference: LOXO-BTK-21050

# INVESTIGATOR AGREEMENT

I have read the protocol and agree to conduct the study as described herein.



31A16 2011

Date

2

# STUDY IDENTIFICATION

| Sponsor | Loxo Oncology, Inc. A wholly owned subsidiary of Eli Lilly and Company 701 Gateway Boulevard, Suite 420 South San Francisco, CA 94080 USA Tel (main): (650) 989-8051 |
|---|---|
| Sponsor's Study Contact | PPD Senior Clinical Trial Manager Loxo Oncology, Inc. Tel (mobile): PPD Email: PPD |
| Sponsor's Medical Contact | PPD MD, PhD Medical Monitor, Consulting to Loxo Oncology, Inc. Tel (mobile): PPD Email: PPD |
| Serious Adverse Event Reporting | Email: SAEIntake@labcorp.com |
| Study Site(s) | Coordinating Investigator Study Site Labcorp Clinical Research Unit Inc. 3402 Kinsman Boulevard Madison, WI 53704 USA |
| | Up to 2 additional sites in the United States may be utilized. |
| Coordinating Investigator | PPD MD Labcorp Clinical Research Unit Inc. 3402 Kinsman Boulevard Madison, WI 53704 USA Tel: PPD Tel (after hours): PPD |
| Sub-investigator(s) | Obtain information from Form FDA 1572 |
| Clinical Laboratory(s) | Meriter Laboratories<br>36 South Brooks Street<br>Madison, WI 53715<br>USA |
| | Each additional site will use their local laboratory for safety analyses. |

# CONFIDENTIAL

#### **SYNOPSIS**

# **Study Title**

A Phase I, Open-Label, Randomized, 2-Way Crossover Study to Compare the PK of Pirtobrutinib (LOXO-305) Tablets

# **Objectives and Endpoints**

The primary objective of the study is to assess the relative bioavailability of a pirtobrutinib tablet lot with a slower dissolution profile (test [T]) relative to the pirtobrutinib tablet lot currently used in the clinical setting (reference [R]) following single doses of pirtobrutinib, as assessed by pirtobrutinib pharmacokinetics (PK) in healthy adult subjects.

The secondary objective of the study is to assess the safety and tolerability of single doses of pirtobrutinib when administered as a test tablet lot and a reference tablet lot in healthy adult subjects.

# **Study Design**

This is a Phase 1, open-label, randomized, 2-way crossover study to compare the PK of pirtobrutinib tablets after a single oral dose in healthy adult subjects.

A single oral dose of pirtobrutinib will be administered as test lot tablets (T) or reference lot tablets (R). The 2 treatment sequences will be TR and RT. Subjects will be randomly assigned to 1 of the 2 treatment sequences, according to a randomization scheme issued by Labcorp Drug Development. Up to 28 healthy adult male and female subjects (women of non-childbearing potential only) will be enrolled.

In Treatment T, a single oral dose of 200 mg pirtobrutinib ( $2 \times 100$  mg) as test lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

In Treatment R, a single oral dose of 200 mg pirtobrutinib ( $2 \times 100$  mg) as reference lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

Blood samples for the analysis of plasma concentrations of pirtobrutinib and for future potential and/or exploratory analysis will be collected from predose through 168 hours postdose for Treatment R and Treatment T.

There will be a washout period of 7 days between the doses of pirtobrutinib administered in Treatments R and T.

The start of the study is defined as the date the first subject who is enrolled in the study signs an informed consent form (ICF). Note that enrolled subjects are defined as those subjects who are assigned to receive a dose of study drug; this definition excludes screen failure subjects. Replacement subjects may be enrolled only if deemed necessary by the Sponsor.

Subjects who are determined to be screen failures are permitted to be re-screened if the Investigator (or designee), with agreement from the Sponsor, feels that the subject may meet eligibility criteria upon re-screen. Re-screened subjects will be provided a new subject number. A minimum of 7 days must elapse between date of screen failure and date of re-screening.

To assess their eligibility to enter the study, potential subjects will be screened within 40 days (Days -41 to -2) and be admitted to the Clinical Research Unit (CRU) on Day -1 (Check-in).

Subjects will be confined at the CRU from the time of Check-in (Day -1) until End of Treatment (EOT) on Day 15 upon completion of all PK and safety assessments or Early Termination (ET) if the subject discontinues. Subjects will be dosed on Day 1 and Day 8. A follow-up phone call will occur for all subjects who received at least 1 dose of study drug (including subjects who are terminated early) 7 days ( $\pm$  2 days) after EOT or ET. The duration of participation is expected to be approximately 65 days (Screening through follow-up phone call).

In this study, physical examinations, 12-lead electrocardiograms (ECGs), vital sign measurements, How Do You Feel? (HDYF?) inquiries, clinical chemistry panel, coagulation parameters, hematology panel, urinalysis (Appendix 2), and recording of concomitant medications will be performed at specified times during the study (for specific timepoints and details on each study variable, refer to Appendix 4).

Adverse events (AEs) and serious AEs (SAEs) will be collected beginning at informed consent. Adverse events will be reported throughout the study (ie, from signing of the ICF until End of Study [EOS], or until ET if the subject discontinues from the study and does not complete a follow-up phone call), either as subject medical history (if the event is reported as beginning prior to signing of the ICF or if the event occurs prior to study drug administration on Day 1 and is assessed as not related to study procedures by the Investigator [or designee]) or as AEs (if the event occurs after signing of the ICF but prior to study drug administration on Day 1 and is assessed as related to study procedures by the Investigator [or designee], or if the event occurs after study drug administration on Day 1 through EOT or ET regardless of relationship to study drug). From EOT or ET through EOS, only AEs assessed as related to study drug by the Investigator (or designee) are to be reported. All SAEs that develop from the time of ICF signing until EOS (or ET, if the subject discontinues from the study and does not complete a follow-up phone call) are to be reported.

Study completion is defined as the time of the last subject's follow-up phone call.

# **Number of Subjects**

Up to 28 healthy adult male and female subjects (women of non-childbearing potential only) will be enrolled. Every attempt will be made to enroll at least 3 subjects of each sex in the study.

# Diagnosis and Main Criteria for Inclusion

Male subjects, and female subjects of non-childbearing potential must meet the following criteria:

- Between 18 and 55 years of age, inclusive, at Screening
- Within body mass index range 18.0 to 32.0 kg/m<sup>2</sup>, inclusive
- In good general health, based on medical history, physical examination findings, vital signs, 12-lead ECGs, or clinical laboratory evaluations at Screening and/or Check-in (Day -1), as determined by the Investigator (or designee).

## Investigational Medicinal Products, Dose, and Mode of Administration

Subjects will receive each of the following treatments once throughout the study:

## Treatment T

A single oral dose of 200 mg pirtobrutinib (as  $2 \times 100$  mg) as test lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

#### Treatment R

A single oral dose of 200 mg pirtobrutinib (as  $2 \times 100$  mg) as reference lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

Administration of pirtobrutinib in Treatments T and R (on Day 1 or Day 8) should occur at approximately the same time (±15 minutes). Pirtobrutinib will be administered orally with approximately 240 mL of water. An additional 100 mL of water may be administered if needed.

# **Duration of Subject Participation in the Study**

Planned Enrollment/Screening Duration: Approximately 40 days (Days -41 to -2).

Length of CRU Confinement: Up to 16 days (Days -1 to 15).

Planned Study Conduct Duration: Up to 65 days (Screening through follow-up call).

#### Criteria for Evaluation:

#### **Pharmacokinetics:**

Serial PK blood samples for the analysis of plasma concentrations of pirtobrutinib and for future potential and/or exploratory analysis will be collected from predose through 168 hours post-pirtobrutinib administration in Treatment T and Treatment R.

The following PK parameters will be calculated, whenever possible, based on the plasma concentrations of pirtobrutinib (as appropriate): area under the concentration-time curve (AUC) from hour 0 to 24 hours postdose (AUC<sub>0-24</sub>), AUC from hour 0 to the last measurable concentration (AUC<sub>0-t</sub>), AUC from hour 0 extrapolated to infinity (AUC<sub>0-inf</sub>), percentage extrapolation for AUC<sub>0-inf</sub> (%AUC<sub>extrap</sub>), maximum observed plasma concentration (C<sub>max</sub>), time to C<sub>max</sub> (t<sub>max</sub>), apparent terminal elimination rate constant ( $\lambda_Z$ ), apparent systemic clearance (CL/F), apparent plasma terminal elimination half-life (t<sub>½</sub>), and apparent volume of distribution (V<sub>z</sub>/F).

# Safety:

Safety will be monitored with HDYF? inquiries, clinical laboratory evaluations, vital sign measurements, 12-lead ECGs, and physical examinations.

#### **Statistical Methods**

#### **Pharmacokinetics:**

The primary PK analysis planned for this study is a mixed effect model including planned treatment sequence, period, and actual treatment as fixed effects and subject within planned treatment sequence as a random effect will be used to analyze the natural log-transformed PK parameters (AUC<sub>0-t</sub>, AUC<sub>0-inf</sub>, and C<sub>max</sub>) and will include calculation of least squared (LS) means and the difference between treatment LS means, as well as their corresponding 90% confidence intervals (CIs). The geometric mean ratios and their 90% CIs of the PK parameter for each treatment comparison will be constructed using the exponentiation of the difference and the CIs from the mixed effect model. The comparison of interest is Treatment T (as test) compared with Treatment R (as reference).

#### **Safety:**

All safety assessments, including AEs, SAEs, vital sign measurements, clinical laboratory results, physical examination results, concomitant medications, and 12-lead ECGs, will be tabulated, and summarized where possible, using descriptive methodology by treatment and,

Protocol CONFIDENTIAL Labcorp Drug Development Study: 8478595 Protocol Reference: LOXO-BTK-21050

as needed, by timepoint. Unless otherwise specified, baseline value is defined as the last non-missing measurement before administration of study drug for each period (ie, Day 1 and Day 8). No formal statistical analyses are planned for the safety data. All safety data will be listed by subject.

The specific procedures will be documented in the statistical analysis plan.

# TABLE OF CONTENTS

| TITLE PAGE | 1 |
|----------------------------------------------------------|----|
| INVESTIGATOR AGREEMENT | 3 |
| STUDY IDENTIFICATION | 4 |
| SYNOPSIS | 6 |
| TABLE OF CONTENTS | 11 |
| LIST OF TABLES AND FIGURES | 14 |
| LIST OF ABBREVIATIONS | 15 |
| 1. INTRODUCTION | 16 |
| 1.1. Background | 17 |
| 1.2. Nonclinical Pharmacokinetics and Toxicology Summary | 17 |
| 1.3. Summary of Clinical Experience | 19 |
| 1.3.1. Safety | 21 |
| 1.3.2. Pharmacokinetics | 22 |
| 1.4. Study Rationale | 26 |
| 1.5. Risk Assessment | 26 |
| 2. OBJECTIVES AND ENDPOINTS | 27 |
| 2.1. Objectives | 27 |
| 2.1.1. Primary Objective | 27 |
| 2.1.2. Secondary Objective | 27 |
| 2.2. Endpoints | 27 |
| 2.2.1. Primary Endpoints | 27 |
| 2.2.2. Secondary Endpoints | 27 |
| 3. INVESTIGATIONAL PLAN | 28 |
| 3.1. Overall Study Design and Plan | 28 |
| 3.2. Discussion of Study Design | 30 |
| 3.3. Selection of Doses in the Study | 30 |
| 3.3.1. Pirtobrutinib | 30 |
| 4. SELECTION OF STUDY POPULATION | 30 |
| 4.1. Screening Procedures | 30 |
| 4.2. Check-in Procedures (Day -1) | 31 |
| 4.3. Inclusion Criteria | 32 |
| 4.4. Exclusion Criteria | 34 |
| 4.5. Subject Number and Identification | 37 |
| 4.6. Removal of Subjects from Study Participation | 38 |
| 5. STUDY TREATMENTS | 39 |
| 5.1. Description, Storage, Packaging, and Labeling | 39 |
| 5.2. Study Treatment Administration | 39 |
| 5.1. Randomization | 40 |

| | 5.2. | Blinding | 40 |
|---|---|---|---|
| | 5.3. | Treatment Compliance | 40 |
| | 5.4. | Drug Accountability | 41 |
| 6. | CON | NCOMITANT THERAPIES AND OTHER RESTRICTIONS | 41 |
| | 6.1. | Concomitant Therapies | 41 |
| | 6.2. | Diet, Fluid, and Activity Control | 41 |
| 7. | STU | JDY ASSESSMENTS AND PROCEDURES | 42 |
| | 7.1. | Pharmacokinetic Assessments | 42 |
| | 7. | .1.1. Pharmacokinetic Blood Sample Collection and Processing | g42 |
| | 7. | .1.2. Analytical Methodology | 42 |
| | 7.2. | Safety and Tolerability Assessments | 43 |
| | 7.2 | .2.1. Adverse Events | 43 |
| | 7.2 | .2.2. Clinical Laboratory Evaluations | 44 |
| | 7.2 | .2.3. Vital Signs | 45 |
| | 7.2 | .2.4. 12-lead Electrocardiogram | 45 |
| | 7.2 | .2.5. Physical Examination | 45 |
| 8. | SAM | MPLE SIZE AND DATA ANALYSIS | 45 |
| | 8.1. | Determination of Sample Size | 45 |
| | 8.2. | Analysis Populations | 46 |
| | 8.2 | .2.1. Pharmacokinetic Population | 46 |
| | 8.2 | .2.2. Safety Population | 46 |
| | 8.3. | Pharmacokinetic Analysis | 46 |
| | 8.3 | .3.1. Descriptive Analysis | 47 |
| | 8.3 | .3.2. Statistical Methodology | 47 |
| | 8.4. | Safety Analysis | 47 |
| | 8.5. | Data Handling and Record Keeping | 47 |
| | 8.6. | Quality Control and Quality Assurance | 48 |
| 9. | ADN | MINISTRATIVE ASPECTS | 49 |
| | 9.1. | Change in Protocol | 49 |
| | 9.2. | Site Initiation Visit/Investigator Meeting | 49 |
| | 9.3. | Disclosure | 49 |
| | 9.4. | Monitoring | 49 |
| | 9.5. | Institutional Review Board | 50 |
| | 9.6. | Informed Consent | 50 |
| | 9.7. | Records | 50 |
| | 9.8. | Reference to Declaration of Helsinki/Basic Principles | 51 |
| | 9.9. | Financing and Insurance | 51 |
| 10 | . REF | FERENCES | 51 |
| 11 | ΔPP | PENDICES | 52 |

| Protocol | CONFIDENTIAL |
|---|---|
| Labcorp Drug Development Study: 8478595 | Protocol Reference: LOXO-BTK-21050 |
| Appendix 1: Adverse Event Reporting | 53 |
| Appendix 2: Clinical Laboratory Evaluations | |
| Appendix 3: Total Blood Volume | 58 |
| Appendix 4: Schedule of Assessments | 59 |

# LIST OF TABLES AND FIGURES

| Table 1: Clinical Pharmacology Studies | 20 |
|---|---|
| Table 2: Frequency of Treatment-related Treatment-emergent Adverse Events Reported in Clinical Pharmacology Studies | |
| Table 3: Pharmacokinetic Parameters of Pirtobrutinib in Cancer Patients (Study LOXO-BTK-18001) at Steady State (Cycle 1 Day 8) | 24 |
| Table 4: Study Drugs | 39 |
| Figure 1: Arithmetic Mean (± SD) Plasma Concentrations of Pirtobrutinib Following Daily Oral Administrations on Day 1 (top panel) and Day 8 (bottom panel) of Cycle 1 in Cancer Patients | 25 |
| Figure 2: Dose-exposure Correlation Assessed by AUC <sub>0-8</sub> vs Dose for Cycle 1 Day 8 | 26 |
| Figure 3: Study Schematic | 29 |

#### LIST OF ABBREVIATIONS

%AUC<sub>extrap</sub> percentage extrapolation for area under the concentration-time curve

from hour 0 extrapolated to infinity

ADL Activities of Daily Living

AE adverse event

AUC area under the concentration-time curve

 $AUC_{0-24}$  area under the concentration-time curve from hour 0 to 24 hours postdose

AUC<sub>0-inf</sub> area under the concentration-time curve from hour 0 extrapolated to

infinity

 $AUC_{0-t}$  area under the concentration-time curve from hour 0 to the last

measurable concentration

AV atrioventricular BID twice daily

BMI body mass index BP blood pressure

BTK Bruton's tyrosine kinase
CFR Code of Federal Regulations

C-G Cockcroft-Gault
CI confidence interval

CL/F apparent systemic clearance CLL chronic lymphocytic leukemia

C<sub>max</sub> maximum observed plasma concentration

COVID-19 SARs Coronavirus 19
CrCl creatinine clearance
CRU Clinical Research Unit

CTCAE Common Terminology Criteria for Adverse Events

CV coefficient of variation
CYP cytochrome P450
ECG electrocardiogram

eCRF electronic case report form

EOS End of Study
EOT End of Treatment
ET Early Termination

FDA Food and Drug Administration FSH follicle-stimulating hormone GLP good laboratory practice

HbA1c hemoglobin A1c

HBsAg hepatitis B surface antigen

HBV hepatitis B virus
HCV hepatitis C virus
HDYF? How Do You Feel?

hERG human ether-à-go-go-related gene HIV human immunodeficiency virus

HR heart rate

HRT hormone replacement therapy

IB investigator's brochure

IC<sub>50</sub> 50% inhibitory concentration

ICF informed consent form IgM immunoglobulin M

IRB institutional review board

IUD intrauterine device LFT liver function test

LS least squares

NHL non-Hodgkin lymphoma PCR polymerase chain reaction

P-gp P-glycoprotein PK pharmacokinetic

QD once daily

QTc QT interval corrected

QT cF QT interval corrected for heart rate using Fridericia's method

SAE serious adverse event SAP statistical analysis plan

SLL small lymphocytic lymphoma SOP standard operating procedure

SUSAR suspected unexpected serious adverse reaction apparent plasma terminal elimination half-life

TEAE treatment-emergent adverse event

TFLs tables, figures, and listings

time to maximum observed plasma concentration

TSH thyroid-stimulating hormone

UA urinalysis
US United States

 $V_z/F$  apparent volume of distribution WHO World Health Organization

 $\lambda_Z$  apparent terminal elimination rate constant

#### 1. INTRODUCTION

Refer to the investigator's brochure (IB) for detailed information concerning the available pharmacology, toxicology, drug metabolism, clinical studies, and adverse event (AE) profile of the investigational medicinal product, pirtobrutinib.<sup>1</sup>

## 1.1. Background

Pirtobrutinib (also known as LOXO-305 and LY3527727) is a selective inhibitor of the Bruton's tyrosine kinase (BTK) being developed by Loxo Oncology. Pirtobrutinib is distinct from the approved BTK inhibitors (ibrutinib, acalabrutinib, and zanubrutinib) in several important ways including on the basis of its selectivity, favorable absorption, distribution, metabolism, and excretion properties, and non-covalent binding mode.<sup>2</sup> These features enable pirtobrutinib to achieve pharmacokinetic (PK) exposures that exceed the BTK concentration resulting in 90% inhibition at trough, and thus deliver tonic BTK target inhibition throughout the dosing period, regardless of the intrinsic rate of BTK turnover. Moreover, the non-covalent binding mode of pirtobrutinib is unaffected by BTK C481 substitutions, a common mechanism of drug resistance described for all available covalent inhibitors. 3,4,5,6,7 Finally, pirtobrutinib is also a highly selective molecule that is more than 300-fold more selective for BTK versus 370 other kinases tested with no significant inhibition of non-kinase off-targets at 1 µM, thus limiting the potential for off-target mediated toxicities. Collectively, these unique properties of pirtobrutinib are expected to deliver more potent, continuous, and selective inhibition of BTK in a variety of settings, potentially resulting in increased efficacy. Of note, the activity of pirtobrutinib in diverse preclinical model systems supports this underlying hypothesis.<sup>2</sup>

Pirtobrutinib is a small molecule that was designed to block the adenosine triphosphate binding site of the BTK competitively. Pirtobrutinib has a molecular weight of approximately 500 g/mol.

# 1.2. Nonclinical Pharmacokinetics and Toxicology Summary

Pirtobrutinib had high permeability in vitro, but low aqueous solubility. To reduce the variability in oral absorption, a tablet formulation was developed that showed consistent oral bioavailability of approximately 50% in rats and 80% in dogs. The bioavailability of the formulation was also not dependent on feeding state in dogs. Refer to the IB for further details.<sup>1</sup>

As is common in rodents, oral exposure of pirtobrutinib was consistently much higher in female rats than in males given the same dose of pirtobrutinib. The sex difference was also apparent after intravenous administration of pirtobrutinib. There was no difference in the PK of pirtobrutinib between sexes of dog, and none is expected in other non-rodent species, including humans.

The volume of distribution of pirtobrutinib ranged from approximately 2 L/kg in the dog to 5 L/kg in the male rat, which indicates that pirtobrutinib distributes into tissues. Pirtobrutinib had protein binding of approximately 95% in human plasma. A somewhat lower extent of binding (approximately 82% to 92%) was observed across mouse, rat, rabbit, and dog.

Pirtobrutinib was metabolized slowly by human microsomal fractions and hepatocytes. The low rates of metabolism in both these human in vitro systems suggest that pirtobrutinib will have low clearance in humans. In vitro data with clone-expressed cytochrome P450 (CYP) enzymes and human liver microsomes indicate that CYP3A4 is the primary CYP enzyme that metabolizes pirtobrutinib.

In long-term hepatocyte incubations, pirtobrutinib was metabolized by both oxidation and glucuronidation. Inhibition of oxidative metabolism by addition of the P450 inhibitor 1-aminobenzotriazole showed that oxidative metabolism is CYP dependent. All metabolites formed by human hepatocytes were also formed in rat and/or dog hepatocytes supporting the use of rat and dog for nonclinical safety assessment.

Renal clearance of pirtobrutinib in male and female rats was negligible. No data on renal clearance are available in other species; however, the renal excretion pathway is often conserved across species, and therefore no renal clearance would be expected in humans.

In a good laboratory practice (GLP) in vitro assay for human ether-à-go-go-related gene (hERG) activity, the concentration resulting in 50% inhibitory concentration (IC<sub>50</sub>) for the inhibitory effects of pirtobrutinib on hERG potassium currents was uM, which is approximately **CC** higher than the maximum unbound concentration of pirtobrutinib in patients treated with the dose of 200 mg once daily (QD). There were no pirtobrutinib-related changes in any cardiovascular endpoints including QT interval corrected (QTc) at single doses up to 60 mg/kg in the GLP cardiovascular study in the conscious telemetry-instrumented dog. The maximum observed plasma concentration (C<sub>max</sub>) for this dose was CCI ng/mL, which is approximately CCI above the predicted C<sub>max</sub> (CCI ng/mL) at the proposed clinical therapeutic dose of 200 mg QD. Furthermore, there were no pirtobrutinib-related abnormalities in rhythm or waveform morphology in the GLP 28-day repeated-dose toxicity study in dogs at the low and mid-dose groups based on comparison of predose and postdose electrocardiogram (ECG) recordings. The high dose (90/60 mg/kg/dose twice daily [BID]) was not evaluated as animals in this group were moribund/debilitated and were terminated on Day 13. Mean QTc interval was statistically significantly prolonged (+6%; +15 msec) on Day 26 of the dosing phase in males administered 30/10 mg/kg/dose BID compared with controls. The prolongation in QTc for males was below the 10% increase or the threshold reported for canines exposed to therapeutic concentrations of drugs known to cause QT prolongation in humans. 8 Therefore, the QTc changes were considered physiologically unimportant, and thus not deemed to be adverse. Together, these data indicate that pirtobrutinib has a low risk of inducing delayed ventricular repolarization, prolongation of the QTc interval, and unstable arrhythmias in patients.

There were no pirtobrutinib-related findings on the central nervous system when evaluated in rat-functional observational battery tests and locomotor activity assessments after 4 weeks of dosing or during recovery at doses of up to 500 mg/kg/dose BID in male rats and 175 mg/kg/dose BID in female rats as part of the GLP 28-day repeat-dose study.

Pirtobrutinib had no effect on respiration rate in the dog at doses up to 10 mg/kg/dose BID.

Targets of toxicity were characterized in repeated-dose studies conducted in 2 relevant toxicity species. Certain targets (the hematopoietic and lymphoid systems) were found in both the rat and the dog. Rat-specific changes in the pancreas are species-specific and seen with other BTK inhibitors. Dog-specific changes in lung and large intestine were lesions contributing to moribundity in high-dose animals in the 28-day study. Doses evaluated in the 28-day dog study demonstrated a steep dose-response curve for toxicity and pronounced changes in hematologic parameters at high exposures. Additionally, in dogs treated for

3 months, 2 male dogs at 5 mg/kg BID (the highest dose tested) were observed to have eye lesions via both ophthalmic and microscopic examination. Findings were observed in both eyes of these animals and consisted of very slight to slight multifocal or focal areas of corneal opacity in the center of the cornea along with constellation histopathological findings suggestive of minimal to mild corneal injury. The time of onset of these effects is unknown, as ophthalmic exams were only performed prior to the start of dosing and during the last week of the study; however, no eye effects were observed in the previous 28-day study. No ocular findings were observed in females. See the IB for additional details.<sup>1</sup>

Pirtobrutinib was not mutagenic in 2 bacterial reverse mutation assays and was negative in a non-GLP micronucleus assay using Chinese hamster ovary cells. Pirtobrutinib was positive for the induction of micronuclei via an aneugenic mechanism in the absence and presence of the exogenous metabolic activation system in a GLP in vitro micronucleus assay in human peripheral blood lymphocytes. However, pirtobrutinib was negative in a GLP in vivo micronucleus assay in rats at doses up to and including a dose of the Communication of the Communication of the communication of the

Pirtobrutinib was not found to be phototoxic when evaluated in an in vitro neutral red uptake phototoxicity assay.

# 1.3. Summary of Clinical Experience

The summary of clinical experience is based on data generated from studies conducted using a reference pirtobrutinib tablet. Pirtobrutinib is currently being studied in an ongoing global Phase 1/2 first-in-human study, LOXO-BTK-18001 (the BRUIN study), in patients with previously treated chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) or non-Hodgkin lymphoma (NHL). Pirtobrutinib is also being studied in one Phase 2 study and three Phase 3 studies in patients with hematological malignancies. In addition, pirtobrutinib has been investigated in 12 clinical pharmacology studies, 1 of which is ongoing (Table 1).

The safety and PK data are summarized in Sections 1.3.1 and 1.3.2. At the time of this protocol's development, no safety or PK data is available from the Phase 2/3 studies.

Protocol CONFIDENTIAL Labcorp Drug Development Study: 8478595 Protocol Reference: LOXO-BTK-21050

**Table 1: Clinical Pharmacology Studies** 

| Protocol<br>Reference | Brief Study Title | Dosing<br>Regimen | Study Status | Actual<br>Enrollment |
|---|---|---|---|---|
| LOXO-BTK-20014 | Pilot study of the effect of food and omeprazole on PK of pirtobrutinib | 200 mg SD | Completed | 10 |
| LOXO-BTK-20009 | Effect of food on PK of pirtobrutinib | 200 mg SD | Closed to enrollment; CSR pending | 20 |
| LOXO-BTK-20007 | DXO-BTK-20007 Metabolism study of an oral dose of [14C]-pirtobrutinib and IV microtracer dose of [14C]-pirtobrutinib given at t <sub>max</sub> of an oral dose of non-labelled pirtobrutinib | | Closed to<br>enrollment;<br>CSR pending | 9 |
| 6 8 | | 300 mg;<br>600 mg;<br>800 mg;<br>900 mg SD | Completed | 24 |
| | | 200 mg QD;<br>13 days | Completed | 15 |
| LOXO-BTK-20006 | XO-BTK-20006 DDI of the effect of itraconazole and rifampin on the PK of pirtobrutinib | | Completed | 27 |
| LOXO-BTK-20016 | OXO-BTK-20016 DDI of the effect of pirtobrutinib on the PK of repaglinide | | Completed | 16 |
| LOXO-BTK-20010 DDI of the effect of pirtobrutinib on the PK of a sensitive CYP1A2, CYP2C9, and CYP2C19 substrate (cocktail study) | | 200 mg QD;<br>14 days | Closed to enrollment; CSR pending | 16 |
| LOXO-BTK-20021 DDI of the effect of pirtobrutinib on the PK of a P-gp transporter substrate digoxin | | 200 mg QD;<br>9 days | Closed to enrollment; CSR pending | 16 |
| LOXO-BTK-20011 Evaluation of potential for QT prolongation by pirtobrutinib | | 900 mg SD | Closed to enrollment; CSR pending | 31 |
| LOXO-BTK-20013 Study of pirtobrutinib in subjects with mild, moderate, and severe renal impairment disease versus matched healthy controls* | | 200 mg SD | Closed to enrollment; CSR pending | 16 |
| LOXO-BTK-20012 Study of pirtobrutinib in subjects with mild, moderate, and severe hepatic impairment versus matched healthy controls | | 200 mg SD | Enrolling | 24* |

Abbreviations: CSR = clinical study report; CYP = cytochrome P450; DDI = drug-drug interaction; IV = intravenous; P-gp = P-glycoprotein; PK = pharmacokinetic; QD = once daily; SD = single dose; t<sub>max</sub> = time to maximum observed plasma concentration.

<sup>\*</sup>At the time of this protocol's development, 24 patients had been enrolled.

# **1.3.1.** Safety

The summary of safety information is based on data generated from studies conducted using a reference pirtobrutinib tablet. As of September 27, 2020, 330 patients were treated in the LOXO-BTK-18001 study and received pirtobrutinib. This includes 324 patients treated at doses ranging from 25 mg QD to 300 mg QD in Phase 1/2 Monotherapy cohorts, and 6 patients treated in Phase 1b Combination Arm A (pirtobrutinib 200 mg QD plus venetoclax 400 mg QD [after venetoclax ramp-up]). A full summary of treatment-emergent AEs (TEAEs) for patients in the study is provided in the pirtobrutinib IB and the Investigator is directed to the safety information described in that document. A summary of safety for pirtobrutinib given as monotherapy to patients in the LOXO-BTK-18001 study is provided below:

• In the 324 patients in the Phase 1/2 Monotherapy cohorts, TEAEs reported in ≥ 10% of patients (n = 33 or more) were fatigue (20.1% total, 8.3% related), diarrhea (17.0% total, 8.6% related), and contusion (13.0% total, 9.0% related). Drug-related TEAEs were reported in 156 of 324 patients (48.1%) in the Phase 1/2 Monotherapy cohorts. The most frequently reported drug-related TEAEs for pirtobrutinib (those in > 5% of patients overall) were contusion (9.0%), diarrhea (8.6%), and fatigue (8.3%). All other drug-related TEAEs were reported in < 5% of patients (ie, < 17 patients each). Treatment-emergent AEs of severity Grade 3 or 4 were reported in 87 of 324 patients (26.9%) in the Phase 1/2 Monotherapy cohorts, with 41 (12.7%) of these Grade 3 or 4 AEs reported as related to study drug.

On-study death (death within 28 days of the last dose of study drug) due to a Grade 5 (fatal) AE was reported in 4 of 324 patients (1.2%) in the Phase 1/2 Monotherapy cohorts. One Grade 5 AE, *Enterococcus faecium*-related septic shock, was considered to be related to study drug (further details are provided in the pirtobrutinib IB<sup>1</sup>). All other Grade 5 AEs were considered to be not related to study drug; these included pneumonia fungal, shock, and pleural effusion.

Treatment-related TEAEs have been reported in 30 healthy subjects and 1 subject with severe renal impairment in LOXO-BTK-20014, LOXO-BTK-20006, LOXO-BTK-20017, LOXO-BTK-20007, LOXO-BTK-20008, LOXO-BTK-20016, LOXO-BTK-20011, LOXO-BTK-20010, LOXO-BTK-20009, LOXO-BTK-20021, and LOXO-BTK-20010 (see Table 2). All AEs resolved by the End of Study (EOS).

Protocol CONFIDENTIAL Labcorp Drug Development Study: 8478595 Protocol Reference: LOXO-BTK-21050

Table 2: Frequency of Treatment-related Treatment-emergent Adverse Events Reported in Clinical Pharmacology Studies

| Preferred Term | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5 |
|----------------------|---------|---------|---------|---------|------------|
| Petechiae | 12 | - | - | - | - |
| Headache | 10 | - | - | - | - |
| Diarrhoea | 2 | 1* | - | - | <b>†</b> - |
| Vomiting | 3 | - | - | - | 1- |
| Constipation | 2 | - | - | - | - |
| Abdominal pain upper | 1 | - | - | - | - |
| Feeling abnormal | 1 | - | - | - | - |
| Muscle spasms | 1 | - | - | - | - |
| Flatulence | 1 | - | - | - | - |
| Pollakiuria | 1 | - | - | - | - |
| Dizziness | 1 | - | - | - | - |
| Dysgeusia | 1 | - | - | - | - |
| Dry mouth | 1 | - | - | - | - |
| Abdominal distension | 1 | - | - | - | - |
| Nausea | 1 | - | - | - | - |
| Abdominal discomfort | 1 | - | - | - | - |
| Eructation | 1 | - | - | - | - |

Data are based on both preliminary and final data on file at the time of protocol development.

There have been 3 TEAEs (headache, constipation, diarrhoea) reported following pirtobrutinib administration in healthy volunteers and volunteers with varying degrees of hepatic impairment in the LOXO-BTK-20012 study to date (preliminary data on file at the time of this protocol's development). All TEAEs were Grade 1 (mild) in severity and resolved.

As part of each clinical trial conducted in patients or healthy volunteers, ECG and vital signs are performed at intervals specified by the protocol. For study LOXO-BTK-18001 conducted in patients, no clinically significant findings of QTc prolongation have been identified in 330 patients as of September 27, 2020. In addition, there have been no clinically significant abnormal findings in vital signs and ECG data in the studies investigating pirtobrutinib conducted in healthy volunteers as of the date of this protocol (preliminary data on file at the time of this protocol's development).

#### 1.3.2. Pharmacokinetics

The summary of information is based on data generated from studies conducted using a reference pirtobrutinib tablet. As of September 30, 2020, PK data were available from 181 patients enrolled in the LOXO-BTK-18001 study. Steady-state PK parameters of

<sup>\*</sup>Grade 2 diarrhoea experienced by a subject with severe renal impairment following a single 200-mg dose of pirtobrutinib.

pirtobrutinib in these cancer patients could be derived from data collected on Cycle 1 Day 8 (Figure 1), and are shown in Table 3. These data show that pirtobrutinib is absorbed after oral administration with a median time to maximum observed plasma concentration ( $t_{max}$ ) of approximately 2 hours and low clearance (Table 3). Due to the limited sampling interval (0 to 8 hours), imputation for the 24-hour sample was made from Cycle 1 Day 8 predose sample, leading to an estimated plasma half-life of approximately 20 hours. Maximum observed plasma concentration and area under the plasma concentration-time curve (AUC) of pirtobrutinib showed an increase proportional to dose (Figure 2). Following administration of the recommended Phase 2 dose 200 mg QD, mean trough plasma levels of pirtobrutinib exceeded the concentration required for 96% inhibition of BTK in vitro ( $IC_{50}$  =  $IC_{50}$  |  $IC_{$ 

Pharmacokinetic data following oral administration of a 200-mg dose of pirtobrutinib in tablet form in healthy volunteers in the LOXO-BTK-20014 study indicate that there was little effect of either a standard meal or the proton pump inhibitor (omeprazole) on the PK of pirtobrutinib.

Table 3: Pharmacokinetic Parameters of Pirtobrutinib in Cancer Patients (Study LOXO-BTK-18001) at Steady State (Cycle 1 Day 8)



Abbreviations:

 $AUC_{0-24} = area$  $C_{max} = maximu$ 

of subjects; QD = once daily;  $t_{1/2}$  = half-life;  $t_{max}$  = time of maximal plasma concentration.

 $^{a}$  N = 4,  $^{b}$  N = 5,  $^{c}$  N = 8,  $^{d}$  N = 18,  $^{e}$  N = 64,  $^{f}$  N = 21,  $^{g}$  N = 16,  $^{h}$  N = 73

SDTM Transfer: September 30, 2020







optimization of the commercial site process, differences in the dissolution profiles were identified. Therefore, this study is designed to compare the PK of T2 tablets manufactured at the clinical trial site (reference [R]) and T2 tablets manufactured at the commercial site (test [T]) in healthy subjects.

#### 1.5. Risk Assessment

Subjects in the current study will not receive any health benefit (beyond that of an assessment of their medical status) from participating in the study. The risks of participation are primarily those associated with adverse reactions to the study treatments, although there may also be some discomfort from collection of blood samples and other study procedures. The dose of pirtobrutinib administered in this study is not anticipated to induce any potential risk to subjects participating in this study as the dose does not exceed the highest dose safely administered in first-in-human study or healthy volunteer studies. More information about the known and expected benefits, risks, and reasonably anticipated AEs associated with pirtobrutinib may be found in the IB. I

The safety monitoring practices employed will include AE reporting, vital sign measurements, 12-lead ECGs, clinical laboratory evaluations, and physical examinations, and are considered adequate to protect the subjects' safety.

#### 2. OBJECTIVES AND ENDPOINTS

# 2.1. Objectives

# 2.1.1. Primary Objective

The primary objective of the study is to assess the relative bioavailability of a pirtobrutinib tablet lot with a slower dissolution profile (T) relative to the pirtobrutinib tablet lot currently used in the clinical setting (R) following single doses of pirtobrutinib, as assessed by pirtobrutinib PK in healthy adult subjects.

# 2.1.2. Secondary Objective

The secondary objective of the study is to assess the safety and tolerability of single doses of pirtobrutinib when administered as a test tablet lot and a reference tablet lot in healthy adult subjects.

# 2.2. Endpoints

# 2.2.1. Primary Endpoints

The following PK parameters will be calculated, whenever possible, based on the plasma concentrations of pirtobrutinib (as appropriate):

- AUC from hour 0 to 24 hours postdose (AUC<sub>0-24</sub>)
- AUC from hour 0 to the last measurable concentration (AUC<sub>0-t</sub>)
- AUC from hour 0 extrapolated to infinity (AUC<sub>0-inf</sub>)
- percentage extrapolation for AUC<sub>0-inf</sub> (%AUC<sub>extrap</sub>)
- apparent systemic clearance (CL/F)
- apparent plasma terminal elimination half-life  $(t_{1/2})$
- C<sub>max</sub>
- t<sub>max</sub>
- apparent terminal elimination rate constant  $(\lambda_z)$
- apparent volume of distribution at the terminal phase  $(V_z/F)$

# 2.2.2. Secondary Endpoints

Safety and tolerability will be assessed by monitoring AEs, performing physical examinations and clinical laboratory evaluations, measuring vital signs, and recording 12-lead ECGs.

#### 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design and Plan

This is a Phase 1, open-label, randomized, 2-way crossover study to compare the PK of 2 different lots of pirtobrutinib after a single oral dose in healthy adult subjects.

A single oral dose of pirtobrutinib will be administered as test lot tablets (T2-L [T]) or reference lot tablets (T2-PR [R]). The 2 treatment sequences will be TR and RT. Subjects will be randomly assigned to 1 of the 2 treatment sequences, according to a randomization scheme issued by Labcorp Drug Development. Up to 28 healthy adult male and female subjects (women of non-childbearing potential only) will be enrolled. Replacement subjects may be enrolled only if deemed necessary by the Sponsor. Every attempt will be made to enroll at least 3 subjects of each sex in the study.

In Treatment T, a single oral dose of 200 mg pirtobrutinib ( $2 \times 100$  mg) as test lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

In Treatment R, a single oral dose of 200 mg pirtobrutinib ( $2 \times 100$  mg) as reference lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

Blood samples for the analysis of plasma concentrations of pirtobrutinib and for future potential and/or exploratory analysis will be collected from predose through 168 hours postdose for Treatment R and Treatment T.

There will be a washout period of 7 days between the doses of pirtobrutinib administered in Treatments R and T.

The schematic of the study design is displayed in Figure 3. The start of the study is defined as the date the first subject who is enrolled in the study signs an informed consent form (ICF). Note that enrolled subjects are defined as those subjects who are assigned to receive a dose of study drug; this definition excludes screen failure subjects. Replacement subjects may be enrolled only if deemed necessary by the Sponsor.

Subjects who are determined to be screen failures are permitted to be re-screened if the Investigator (or designee), with agreement from the Sponsor, feels that the subject may meet eligibility criteria upon re-screen. Re-screened subjects will be provided a new subject number. A minimum of 7 days must elapse between date of screen failure and date of re-screening.

To assess their eligibility to enter the study, potential subjects will be screened within 40 days (Days -41 to -2) and be admitted to the Clinical Research Unit (CRU) on Day -1 (Check-in).

Subjects will be confined at the CRU from the time of Check-in (Day -1) until End of Treatment (EOT) on Day 15 upon completion of all PK and safety assessments or Early Termination (ET) if the subject discontinues. Subjects will be dosed on Day 1 and Day 8. A follow-up phone call will occur for all subjects who received at least 1 dose of study drug (including subjects who are terminated early) 7 days (± 2 days) after EOT or ET. The duration of participation is expected to be approximately 65 days (Screening through follow-up phone call).

Screening Period 1 Period 2 Follow-up 7 (± 2) days Days -41 to -2 Day -1 Days 1 to 7 Days 8 to 15 after Discharge Day 1 Day 8 Day 15 Treatment R or Treatment R or Clinic Discharge Treatment T Treatment T EOT/ET PK Sampling: PK Sampling:

Figure 3: Study Schematic

Abbreviations: EOT = End of Treatment; ET = Early Termination; ICF = Informed Consent Form; PK = pharmacokinetic.

Day 1: Predose through

168 hours postdose

Safety Assessments: From signing the ICF to follow-up phone call

Day 8: Predose through

168 hours postdose

In this study, physical examinations, 12-lead ECGs, vital sign measurements, How Do You Feel? (HDYF?) inquiries, clinical chemistry panel, coagulation parameters, hematology panel, urinalysis (UA; Appendix 2), and recording of concomitant medications will be performed at specified times during the study (for specific timepoints and details on each study variable, refer to Appendix 4).

Adverse events and serious AEs (SAEs) will be collected beginning at informed consent. Adverse events will be reported throughout the study (ie, from signing of the ICF until EOS, or until ET if the subject discontinues from the study and does not complete a follow-up phone call), either as subject medical history (if the event is reported as beginning prior to signing of the ICF or if the event occurs prior to study drug administration on Day 1 and is assessed as not related to study procedures by the Investigator [or designee]) or as AEs (if the event occurs after signing of the ICF but prior to study drug administration on Day 1 and is assessed as related to study procedures by the Investigator [or designee], or if the event occurs after study drug administration on Day 1 through EOT or ET regardless of relationship to study drug). From EOT or ET through EOS, only AEs assessed as related to study drug by the Investigator (or designee) are to be reported. All SAEs that develop from the time of ICF signing until EOS (or ET, if the subject discontinues from the study and does not complete a follow-up phone call) are to be reported.

A Schedule of Assessments is presented in Appendix 4. Study completion is defined as the time of the last subject's follow-up phone call.

## 3.2. Discussion of Study Design

Subjects will be randomized to 1 of the 2 treatment sequences to minimize assignment bias. The 2 treatment sequences will be RT and TR. Subjects will be randomly assigned to 1 of the 2 treatment sequences, according to the randomization scheme issued by Labcorp Drug Development. A crossover design is used to reduce the residual variability as every subject acts as their own control. The washout period of 7 days between pirtobrutinib doses in Treatments R and T is considered sufficient to prevent carryover effects of the treatments (greater than 5 half-lives for pirtobrutinib). This study will be open label because the primary endpoints are not considered subjective.

Conducting the study in healthy adult subjects mitigates the potential confounding effects of the disease state and concomitant medications.

# 3.3. Selection of Doses in the Study

#### 3.3.1. Pirtobrutinib

A single oral dose of 200 mg pirtobrutinib will be evaluated as this dose level given QD has been chosen as the recommended Phase 2 dose for the ongoing global Phase 1/2 first-in-human study, LOXO-BTK-18001 in patients with previously treated CLL/SLL or NHL. The available data demonstrate that pirtobrutinib appears safe and well tolerated at these doses. At all evaluated doses, no dose-limiting toxicities have been identified in humans.<sup>1</sup>

#### 4. SELECTION OF STUDY POPULATION

# 4.1. Screening Procedures

The following screening procedures will be performed for all potential subjects at a visit conducted within 40 days of study entry (ie, prior to Check-in [Day -1]):

- 1. Inclusion/exclusion criteria
- 2. Informed consent
- 3. Demographic data
- 4. Medical history (including review of medication[s])
- 5. Height, weight, and body mass index (BMI)
- 6. 12-lead ECG measured after the subject has been resting in the supine position for at least 10 minutes (Section 7.2.4)
- 7. Vital sign measurements (including body temperature, respiratory rate, oxygen saturation, and supine blood pressure [BP] and pulse rate [measured after the subject has been supine for at least 5 minutes]; Section 7.2.3)
- 8. HDYF? inquiry, AE, SAE, and concomitant medication evaluations (Section 7.2.1)
- 9. Clinical laboratory evaluations (Section 7.2.2; clinical chemistry panel [fasted at least 8 hours], coagulation parameters, hematology panel, and UA; Appendix 2)

Protocol Reference: LOXO-BTK-21050

- 10. Screens for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), hepatitis B virus (HBV) immunoglobulin M (IgM) core antibody, human immunodeficiency virus (HIV) antibody, and SARs Coronavirus 19 (COVID-19) via polymerase chain reaction (PCR) testing or equivalent (Appendix 2)
- 11. Hemoglobin A1c (HbA1c) test (Appendix 2)
- 12. Urine drug screen for selected drugs of abuse (including cotinine) and alcohol screen (breath or urine; Appendix 2)
- 13. Creatinine clearance (CrCl) calculated using the Cockcroft-Gault (C-G) equation (Appendix 2)
- 14. Pregnancy test (for female subjects only; Appendix 2)
- 15. Follicle-stimulating hormone (FSH) test (for post-menopausal female subjects only; Appendix 2)
- 16. Thyroid-stimulating hormone (TSH) test (Appendix 2).

# 4.2. Check-in Procedures (Day -1)

At Check-in (Day -1), subjects will report to the CRU and the following procedures will be performed:

- 1. Review of inclusion/exclusion criteria
- 2. Interim medical history, including concomitant medication(s)
- 3. Weight
- 4. Complete physical examination (Section 7.2.5)
- 5. 12-lead ECG measured after the subject has been resting in the supine position for at least 10 minutes (Section 7.2.4)
- 6. Vital sign measurements (including body temperature, respiratory rate, oxygen saturation, and supine BP and pulse rate [measured after the subject has been supine for at least 5 minutes]; Section 7.2.3)
- 7. HDYF? inquiry, AE, SAE, and concomitant medication evaluations (Section 7.2.1)
- 8. Clinical laboratory evaluations (Section 7.2.2; clinical chemistry panel [fasted at least 8 hours], coagulation parameters, hematology panel, and UA; Appendix 2)
- 9. Screen for COVID-19 via PCR test (or equivalent; Appendix 2)
- 10. Urine drug screen for selected drugs of abuse (including cotinine) and alcohol screen (breath or urine; Appendix 2)
- 11. CrCl calculated using the C-G equation (Appendix 2)
- 12. Pregnancy test (for female subjects only; Appendix 2)
- 13. Compliance with concomitant medications and exclusionary restrictions (Section 6).

For subjects to continue their participation in the study, the inclusion/exclusion criteria must continue to be met at Check-in (Day -1 [as appropriate; #1, Section 4.2]). In addition, continued compliance with concomitant medication and other restrictions will be verified.

The Sponsor will review medical history and all screening evaluations for potential subjects prior to Check-in (Day -1). Prior to dosing, the Sponsor will provide approval of subjects selected for enrollment by the Investigator (or designee).

Subjects who meet all the inclusion criteria and for whom none of the exclusion criteria apply will be eligible to be enrolled into the study. Safety evaluations may be repeated at the discretion of the Investigator (or designee) or Sponsor.

#### 4.3. Inclusion Criteria

Subjects who meet the following criteria at Screening and Check-in (Day -1), unless otherwise specified, may be included in the study:

- 1. Males, and females of non-childbearing potential, between 18 and 55 years of age, inclusive, at Screening.
- 2. Within BMI range 18.0 to 32.0 kg/m<sup>2</sup>, inclusive.
- 3. In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital sign measurements, or clinical laboratory evaluations (Appendix 4) at Screening and/or Check-in (Day -1) as assessed by the Investigator (or designee).
- 4. Female subjects of non-childbearing potential, defined as being permanently sterile (ie, due to hysterectomy, bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy, or confirmed tubal occlusion more than 6 months prior to Day 1) or post-menopausal (defined as at least 12 months post-cessation of menses without an alternative medical cause). Post-menopausal status will be confirmed with a screening serum FSH level consistent with post-menopausal status per the laboratory's reference ranges. All female subjects must have a negative qualitative serum or negative qualitative urine pregnancy test (serum human chorionic gonadotropin; quantitative serum human chorionic gonadotropin tests may be used for confirmation as needed and post-menopausal subjects may be eligible for participation if the results of the qualitative serum pregnancy or qualitative urine pregnancy test are positive but the quantitative serum human chorionic gonadotropin results are within the laboratory's reference ranges for post-menopausal women) at Screening and Check-in (Day -1). Female subjects are required to refrain from donation of ova from Check-in (Day -1) until 6 months after Day 8 (or last administration of study drug if subject terminates from the study early).
- 5. Male subjects who are capable of fathering a child must agree to use 1 of the following methods of contraception:
  - a. Male sterilization, with documented confirmation of surgical success. Male subjects will be surgically sterile for at least 90 days prior to Check-in (Day -1), or

Protocol Reference: LOXO-BTK-21050

- b. If documentation of surgical sterilization is not available, male subjects must follow 1 of the contraception methods below from Day 1 through 6 months after Day 8 (or last administration of study drug if subject terminates from the study early):
  - i. Male condom with spermicide, or
  - ii. A male subject must ensure that their female partner meets 1 of the following criteria:
    - 1. intrauterine device (IUD) (hormonal IUD; eg, Mirena<sup>®</sup>). Copper IUDs are acceptable (eg, ParaGard<sup>®</sup>); or
    - 2. established use of oral, implanted, injected, transdermal, intravaginal, or hormonal method of contraception associated with inhibition of ovulation; or
    - 3. non-childbearing potential, defined as being permanently sterile (ie, due to hysterectomy, bilateral tubal ligation, bilateral salpingectomy, bilateral oophorectomy, or confirmed tubal occlusion more than 6 months prior to Day 1 for male partner); or
    - 4. be post-menopausal with amenorrhea for at least 1 year prior to Day 1.

Male subjects who practice true abstinence because of a lifestyle choice (ie, do not become abstinent just for the purpose of study participation) are exempt from contraceptive requirements. Periodic abstinence by a female partner (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. If a male subject is abstinent at the time of signing the ICF but becomes sexually active from Check-in (Day -1) through 6 months after Day 8 (or last administration of study drug if subject terminates from the study early), he must agree to use contraception as described above.

For male subjects, sexual intercourse with female partners who are pregnant, or breastfeeding should be avoided from Check-in (Day -1) through 6 months after Day 8 (or last administration of study drug if subject terminates from the study early), unless the male subject uses a condom with spermicide. Male subjects are required to refrain from donation of sperm from Check-in (Day -1) until 6 months after Day 8 (or last administration of study drug if subject terminates from the study early).

For subjects who are exclusively in same-sex relationships, contraceptive requirements do not apply.

- 6. Able to understand and provide written informed consent.
- 7. Able to comply with all study procedures, including the 15-night stay at the CRU and follow-up phone call.

#### 4.4. Exclusion Criteria

The following will exclude potential subjects from the study:

- 1. History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:
  - a. liver disease
  - b. pancreatitis
  - c. peptic ulcer disease
  - d. intestinal malabsorption
  - e. cholecystectomy
  - f. gastric reduction surgery
  - g. history or presence of clinically significant cardiovascular disease:
    - i. myocardial infarction or cerebrovascular thromboembolism within 6 months prior to Day 1
    - ii. symptomatic angina pectoris within 6 months prior to Day 1
    - iii. congestive heart failure ≥ stage 2 per New York Heart Association Classification within 6 months prior to Day 1
    - iv. congenital prolonged QT syndrome
    - v. ventricular pre-excitation syndrome (Wolff-Parkinson White syndrome)
    - vi. arrhythmia (excluding benign sinus arrhythmia) or history of arrhythmia requiring medical intervention within 6 months prior to Day 1
    - vii. ventricular dysfunction including ventricular fibrillation or risk factors for Torsades de Pointes (eg, heart failure, cardiomyopathy, family history of Long QT Syndrome)
    - viii. ECG abnormalities that are clinically significant at Screening, Check-in (Day -1), or predose on Day 1, including, but not limited to:
      - 1. complete left bundle-branch block
      - 2. first or second-degree atrioventricular (AV) block, type 2, or third-degree AV block
      - 3. QT interval corrected for heart rate (HR) using Fridericia's method (QTcF) > 450 msec

Subjects with out-of-range ECG values or abnormal ECG findings that are not clinically significant will be permitted to have ECGs repeated up to 2 times during Screening, Check-in (Day -1), and predose on Day 1 to confirm eligibility for study

participation, if the repeat value(s) are normal/fall outside of the ranges stated above.

- 2. Subjects with out-of-range, at-rest (ie, supine for at least 5 minutes) vital sign measurements at Screening, Check-in (Day -1), or prior to dosing on Day 1. Out-of-range vital sign measurements are defined as:
  - a. body temperature > 37.5°C;
  - b. pulse rate < 50 or > 99 beats per minute (bpm);
  - c. systolic BP < 89 or > 139 mmHg;
  - d. diastolic BP < 50 or > 89 mmHg;
  - e. oxygen saturation < 95% (room air).

Subjects with out-of-range values for these parameters that are not clinically significant will be permitted to have vital sign measurements repeated up to 2 times during Screening, Check-in (Day -1), and predose on Day 1 to confirm eligibility for study participation if the repeat value(s) are normal/fall outside of the ranges stated above.

- 3. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator (or designee), or mentally or legally incapacitated or has significant emotional problems at the time of the Screening visit or expected during the conduct of the study.
- 4. Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination at Check-in (Day -1).
- 5. Abnormal laboratory values (hematology panel, UA, clinical chemistry panel [fasted at least 8 hours]) that are clinically significant excluding those further defined in exclusion criteria #6, #7, and #8 at Screening and/or Check-in (Day -1). Subjects with out-of-range clinical laboratory results that are not clinically significant (excluding those further defined in exclusion criteria #6, #7, and #8) may have laboratory assessments repeated at the Investigator (or designee)'s discretion up to 2 times during Screening and Check-in (Day -1) to confirm eligibility for study participation if the repeat value(s) fall within normal ranges or are stabilizing.
- 6. Abnormal liver function tests (LFTs) as defined by aspartate aminotransferase, alanine aminotransferase, and serum (total and direct) bilirubin, as well as amylase, or lipase above the upper limit of the normal range per the laboratory's reference ranges at Screening or Check-in (Day -1). Subjects with out-of-range LFTs, amylase, and lipase values above the upper limit of normal that are not clinically significant will be permitted to have LFTs, amylase, or lipase assessments repeated up to 2 times during Screening and Check-in (Day -1) to confirm eligibility for study participation if the repeat value(s) fall within normal ranges.
- 7. Creatine kinase values above the upper limit of the normal range per the laboratory's reference ranges that are clinically significant at Screening or Check-in (Day -1). Subjects with out-of-range creatine kinase values that are not clinically significant will be permitted to have the creatine kinase assessments repeated up to 2 times
Protocol Reference: LOXO-BTK-21050

- during Screening and Check-in (Day -1) to confirm eligibility for study participation if the repeat value(s) are stable or normalizing.
- 8. Creatinine clearance < 90 mL/minute calculated using the C-G equation at Screening or Check-in (Day -1). Subjects with out-of-range CrCl values that are not clinically significant will be permitted to have CrCl assessments repeated up to 2 times during Screening and Check-in (Day -1) to confirm eligibility for study participation if the repeat value(s) fall above the range stated above.
- 9. Hemoglobin A1c  $\geq$  6.5% at Screening. Subjects with out-of-range HbA1c values that are not clinically significant will be permitted to have HbA1c assessments repeated up to 2 times during Screening to confirm eligibility for study participation if the repeat value(s) fall below the range stated above.
- 10. Positive serologic test for HBsAg, HBV IgM core antibody, HCV antibody, or HIV antibody at Screening. Subjects who are positive for HBV IgM core antibody or HCV antibody require confirmation by PCR before enrollment to detect presence of active virus. Subjects who are HBV core antibody or HCV antibody positive or for whom a PCR is unable to be obtained will not be eligible.
- 11. Positive PCR test (or equivalent) for COVID-19 at Screening or Check-in (Day -1). Further details regarding COVID-19 testing (including procedures for subjects who test positive at any time throughout CRU confinement) are specified in a separate document.
- 12. Significant history or clinical manifestation of any allergic, dermatological, biliary, hepatic, gastrointestinal, renal, metabolic, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or heart failure), neurological, thyroid, or psychiatric disorder (as determined by the Investigator [or designee]), or cancer within the past 5 years (except localized basal cell, squamous, or in situ cancer of the skin). Note: subjects with a history of appendectomy and/or hernia repairs will be acceptable.
- 13. History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator (or designee), would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the subject at undue risk.
- 14. History of a major surgical procedure within 30 days prior to Screening.
- 15. Known ongoing alcohol and/or drug abuse within 2 years prior to Screening, or evidence of such abuse as indicated by the laboratory assays for drugs of abuse (including cotinine and alcohol) conducted during Screening and/or at Check-in (Day -1). Tests for drugs of abuse must be negative at both Screening and Check-in (Day -1).
- 16. Use of tobacco, smoking-cessation products, or products containing nicotine and e-cigarettes (nicotine and non-nicotine), within 3 months prior to Screening and through EOT or ET.
- 17. Use or intention to use any prescription or over-the-counter medications (including but not limited to any moderate or strong CYP3A4 and/or CYP3A5 inhibitors or inducers [including herbal products such as St. John's wort], CYP2C8 substrates,

Protocol Reference: LOXO-BTK-21050

strong P-glycoprotein [P-gp] inhibitors, P-gp substrates, proton pump inhibitors, antacids, H<sub>2</sub>-receptor antagonists, and drugs that prolong QT/QTc interval, vitamin supplements, herbal products, natural or herbal supplements, and hormone-replacement therapy [HRT]) from 14 days prior to Day 1 or 5 half-lives (if known, whichever is longer [except for paracetamol/acetaminophen maximum of 2 g/day for up to 3 consecutive days during the study]) through EOT or ET, unless deemed acceptable by the Investigator (or designee) and Sponsor.

- 18. Consumption of grapefruit/grapefruit juice or Seville oranges or its juice within 7 days prior to Check-in (Day -1) and through EOT or ET.
- 19. Consumption of alcohol-containing foods or beverages or caffeine-containing foods or beverages (including but not limited to teas [including decaffeinated teas], coffees [including decaffeinated coffees], colas [including decaffeinated colas], energy drinks, gum containing caffeine, chocolate, and foods and beverages containing chocolate) within 72 hours prior to Check-in (Day -1) and through EOT or ET.
- 20. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
- 21. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator (or designee), within the 30 days prior to Day 1 and through EOT or ET.
- 22. Participation in any other investigational study drug trial in which receipt of any investigational drug occurs in the past 30 days or 5 half-lives (if known), whichever is longer, prior to Day 1.
- 23. Has previously received pirtobrutinib in any other study investigating pirtobrutinib, within 30 days prior to Day 1.
- 24. Strenuous exercise within 5 days prior to Check-in (Day -1) and through EOT or ET.
- 25. Poor peripheral venous access.
- 26. Donation of blood from 56 days prior to Screening; donation of plasma or platelets from 4 weeks prior to Screening.
- 27. Receipt of blood products within 2 months prior to Check-in (Day -1).
- 28. Subjects who, in the opinion of the Investigator (or designee), should not participate in this study.

## 4.5. Subject Number and Identification

Subject numbers will consist of 6 digits in which the first set of 3 digits will identify the site and the second set of 3 digits will identify the subject (eg, 001-101).

For subjects who are withdrawn by the Investigator (or designee) or voluntarily withdraw prematurely from the study, replacement subjects will be enrolled only if deemed necessary by the Sponsor.

If necessary, as determined by the Sponsor, subjects who fail to complete the treatment or have insufficient PK data may be replaced. Replacement subjects will be assigned a subject

number by adding 200 to the last 3 digits of the subject number for the subject they are replacing (eg, Subject Number 001-301 replaces Subject Number 001-101).

Subjects who are determined to be screen failures are permitted to be re-screened if the Investigator (or designee), with agreement from the Sponsor, feels that the subject may meet eligibility criteria upon re-screen. Re-screened subjects will be provided a new subject number as defined above. A minimum of 7 days must elapse between date of screen failure and date of re-screening.

### 4.6. Removal of Subjects from Study Participation

Subjects will be informed that they are free to withdraw from the study at any time and for any reason. The Investigator (or designee) may remove a subject from the study if, in the Investigator's (or designee's) opinion, it is not in the best interest of the subject to continue the study. Subjects may be withdrawn because of the following:

- change in compliance with inclusion/exclusion criterion that is clinically relevant and affects subject safety
- occurrence of AEs
- occurrence of pregnancy
- non-compliance with study restrictions
- intake of non-permitted concomitant medication that might affect subject safety or study assessments/objectives, etc.

Notification of withdrawal will immediately be made to the Sponsor. In case of withdrawal, efforts will be made to perform all ET assessments (Appendix 4). The date the subject is withdrawn from the study and the reason for withdrawal will be recorded on the subject's electronic case report form (eCRF). All withdrawn subjects with AEs that are assessed as related to study drug and which are ongoing at ET may continue to be followed until the symptoms or value(s) return to normal, or acceptable levels, as judged by the Investigator (or designee) and confirmed by the Sponsor.

The entire study may be discontinued at the discretion of the Investigator (or designee) or Sponsor, based on the occurrence of the following:

- AEs unknown to date with respect to their nature, severity, and/or duration
- increased frequency and/or severity and/or duration of known AEs
- medical or ethical reasons affecting the continued performance of the study
- difficulties in the recruitment of subjects
- cancellation of drug development.

In the event that the study is terminated early, the Sponsor or its designee will provide specific guidance to the CRU regarding the EOS procedures.

#### 5. STUDY TREATMENTS

## 5.1. Description, Storage, Packaging, and Labeling

The Sponsor (or designee) will provide the Investigator (or designee) with adequate quantities of the study drug (Table 4).

**Table 4: Study Drugs** 

| Study Drug | Pirtobrutinib | Pirtobrutinib |
|---|---|---|
| Form <sup>a</sup> | Tablet | Tablet |
| Formulation | Test | Reference |
| Strength | 100 mg | 100 mg |
| Supplier | Loxo Oncology, Inc. | Loxo Oncology, Inc. |
| Manufacturer | Lilly del Caribe, Inc. | Bend Research, Inc. |

<sup>&</sup>lt;sup>a</sup> Specific ingredients/purity will be identified in the Certificate of Analysis (or equivalent) that is supplied with the study drug(s).

The tablets containing 100 mg pirtobrutinib will be supplied by the Sponsor (or designee), along with the batch/lot numbers and Certificate of Analysis. It will be provided in high-density polyethylene bottles and will be stored according to the instructions on the label.

Study drugs will be stored at the CRU in a location that is locked with restricted access.

The bulk drug container and unit dose containers will be labeled in accordance with national laws and regulations. The study drugs will be stored in accordance with the labeling. The study drugs will be transferred from bulk supplies into the subject's dose container by qualified CRU employees. Each unit dose container will be appropriately labeled.

### 5.2. Study Treatment Administration

Subjects will receive each of the following treatments once throughout the study:

#### **Treatment T**

• A single oral dose of 200 mg pirtobrutinib (as 2 × 100 mg) as test lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

## **Treatment R**

• A single oral dose of 200 mg pirtobrutinib (as 2 × 100 mg) as reference lot tablets will be administered in the morning on Day 1 or Day 8 (according to the randomization scheme), following a fast of at least 10 hours prior to and 4 hours after dosing. Water

CONFIDENTIAL

Protocol Reference: LOXO-BTK-21050

will be restricted for 1 hour prior to and 1 hour after dosing with the exception of water administered for dose administration.

Administration of pirtobrutinib in Treatments T and R (on Day 1 or Day 8) should occur at approximately the same time (±15 minutes). Pirtobrutinib will be administered orally with approximately 240 mL of water. An additional 100 mL of water may be administered if needed.

Each unit dose will be prepared by qualified CRU staff.

Appropriate unit dose(s), as described above, will be administered to subjects. Although the timing of events requires that each subject will be administered the appropriate dose at a specific time, the exact dose time of subjects may be staggered to obviate the need to have all subjects on precisely the same study schedule. For each dose, the subject's actual dose time will be recorded in the source documents and transcribed into the eCRF.

Subjects will be instructed not to crush, split, or chew the study drugs.

Subjects will not lay supine for 4 hours following pirtobrutinib dose administration, except as necessitated by the occurrence of an AE(s) and/or study procedure(s).

#### 5.1. Randomization

Subjects will be assigned a unique identification number upon screening. Subjects who complete the study screening assessments and meet all the eligibility criteria will be assigned a unique randomization identification number (in accordance with the requirements in Section 4.5 and the randomization scheme generated by Labcorp Drug Development) prior to the time of the first dose, different from the screening number, and will receive the corresponding product according to the randomization scheme generated by Labcorp Drug Development.

Subjects will receive each treatment (T and R) on 1 occasion. The treatments will be administered on Day 1 (Treatment T or R) and Day 8 (Treatment T or R). The sequences to be used in the randomization will be TR and RT.

### 5.2. Blinding

This is an open-label study.

### 5.3. Treatment Compliance

The following measures will be employed to ensure treatment compliance:

- All doses will be administered under the supervision of suitably qualified CRU staff.
- Immediately after oral dose administration, a visual inspection of the mouth and hands will be performed for each subject.
- At each dose preparation occasion, a predose and postdose inventory of pirtobrutinib will be performed.

#### 5.4. Drug Accountability

The Investigator (or designee) will maintain an accurate record of the receipt of pirtobrutinib tablets received. In addition, an accurate drug disposition record will be kept, specifying the amount dispensed to each subject and the date of dispensing. This drug accountability record will be available for inspection at any time. At the completion of the study, the original drug accountability record will be available for review by the Sponsor upon request.

For each batch of unit doses, the empty used unit dose containers will be discarded upon satisfactory completion of the compliance and accountability procedures. Any unused assembled unit doses will be retained until completion of the study.

At the completion of the study, all unused pirtobrutinib tablets will be disposed of by the CRU, in accordance with the CRU's standard operating procedures (SOPs) and local/state/federal guidelines governing waste disposal of investigational drugs, following the Sponsor's written authorization.

#### 6. CONCOMITANT THERAPIES AND OTHER RESTRICTIONS

### **6.1.** Concomitant Therapies

Paracetamol/acetaminophen (maximum of 2 g/day for up to 3 consecutive days) is an acceptable concomitant medication.

Subjects will refrain from participation in any other investigational study drug trial in which receipt of any investigational drug occurs within 5 half-lives (if known) or 30 days, whichever is longer, prior to Day 1.

All prescription medications and over-the-counter medications including but not limited to: moderate or strong CYP3A4 and/or CYP3A5 inhibitors or inducers (including herbal products such as St. John's wort), CYP2C8 substrates, strong P-gp inhibitors, P-gp substrates, proton pump inhibitors, antacids, H<sub>2</sub>-receptor antagonists, and drugs that prolong QT/QTc interval, herbal products, vitamin supplements, natural or herbal supplements, and HRT are prohibited for 14 days or 5 half-lives (if known; except for paracetamol/acetaminophen as referenced above), whichever is longer, prior to Day 1 and through EOT or ET, unless deemed acceptable by the, Investigator (or designee), and Sponsor. Any medication taken by a subject during the course of the study, including details of its dosage, administration, and the reason for its use, will be documented in the eCRF.

The administration of any concomitant medication during the study is prohibited without prior approval of the Investigator (or designee) and Sponsor, unless its use is deemed necessary in a medical emergency. In this case, the use of the concomitant medication will be reported as soon as is practical

### 6.2. Diet, Fluid, and Activity Control

Subjects are required to refrain from use of tobacco, smoking-cessation products, and nicotine-containing products and e-cigarettes (nicotine and non-nicotine) within 3 months prior to Screening through EOT or ET.

Consumption of foods or beverages containing grapefruit/grapefruit juice or Seville oranges or its juice within 7 days prior to Check-in (Day -1) and through EOT or ET will not be allowed.

Consumption of alcohol-containing foods or beverages or caffeine-containing foods or beverages (including but not limited to teas [including decaffeinated teas], coffees [including decaffeinated coffees], colas [including decaffeinated colas], energy drinks, gum containing caffeine, chocolate, and foods and beverages containing chocolate) within 72 hours prior to Check-in (Day -1) and through EOT or ET will not be allowed.

Subjects will refrain from strenuous exercise from 5 days prior to Check-in (Day -1) and during the period of confinement at the CRU and will otherwise maintain their normal level of physical activity through EOT or ET (ie, should not begin a new exercise program or participate in any unusually strenuous physical exertion).

While confined at the CRU, subjects will receive a standard diet at scheduled times that do not conflict with other study-related activities. All study drugs will be administered orally with approximately 240 mL of water. An additional 100 mL of water may be administered if needed.

Fasting requirements and water restrictions in relation to dosing are described in Section 3.1 and Section 5.2.

#### 7. STUDY ASSESSMENTS AND PROCEDURES

#### 7.1. Pharmacokinetic Assessments

### 7.1.1. Pharmacokinetic Blood Sample Collection and Processing

Blood samples for PK analysis of plasma concentrations of pirtobrutinib and for future potential and/or exploratory analysis will be collected at the timepoints specified in Appendix 4. The exact time of the study drug administration and the actual time of blood sampling for PK analysis and for future potential and/or exploratory analysis will be recorded on the eCRF.

Processing, storage, and shipping instructions for these PK blood samples and for future potential and/or exploratory analysis will be provided in a separate Laboratory Manual. The number of blood samples and total blood volume required for PK and for future potential and/or exploratory analysis is presented in Appendix 3.

### 7.1.2. Analytical Methodology

Plasma concentrations of pirtobrutinib will be determined using validated bioanalytical method. Specifics of the bioanalytical method will be provided in a separate document.

Samples collected for the analysis of plasma concentrations of pirtobrutinib may be stored and analyzed for future exploratory analysis, such as quantification of metabolites of pirtobrutinib.

## 7.2. Safety and Tolerability Assessments

Safety evaluations may be repeated at the discretion of the Investigator (or designee) or Sponsor.

Every effort will be made to schedule and perform the procedures in accordance with the nominal time, giving considerations to appropriate posture conditions, practical restrictions, and any other procedures to be performed at the same timepoint. The order of priority for scheduling procedures around a timepoint is (in order of priority):

- dosing
- PK blood sampling
- vital sign measurements\*
- 12-lead ECGs\*
- blood and urine samples for clinical laboratory evaluations
- physical examination.

\* When vital sign measurements and 12-lead ECGs are scheduled at the same time as PK blood sampling, the PK blood sampling will be obtained at the scheduled timepoint, and the vital sign measurements followed by 12-lead ECGs will be obtained prior to and as close as possible to the scheduled PK blood sampling.

#### **7.2.1.** Adverse Events

Adverse event definitions; assignment of severity, causality, action taken, and outcome; and procedures for reporting SAEs are detailed in Appendix 1.

Subjects will be asked a non-leading HDYF? question such as "Have there been any changes in your health status since Screening/since you were last asked?" at the timepoints specified in Appendix 4 (ie, at Screening [after the ICF is signed], at Check-in [Day -1], at each postdose vital sign measurement, and at an appropriate time for all other days). Subjects will also be encouraged to voluntarily report AEs occurring at any other time through the EOS.

Adverse events, whether volunteered, identified by the subject's responses to HDYF? inquiries, or noted on physical examination, ECG, vital sign measurements, or clinical laboratory evaluations, will be recorded throughout the study (ie, from signing of the ICF until EOS [or ET if the subject discontinues from the study and does not complete a follow-up phone call]), either as subject medical history (if the event is reported as beginning prior to signing of the ICF or if the event occurs prior to study drug administration on Day 1 and is assessed as not related to study procedures by the Investigator [or designee]) or as AEs (if the event occurs after signing of the ICF but prior to study drug administration on Day 1 and is assessed as related to study procedures by the Investigator [or designee], or if the event occurs after study drug administration on Day 1 through EOT or ET regardless of relationship to study drug). From EOT or ET through EOS, only AEs assessed as related to study drug by the Investigator (or designee) are to be reported. All SAEs that develop from the time of ICF

signing until EOS (or ET, if the subject discontinues from the study and does not complete a follow-up phone call) are to be reported.

Unless a subject withdraws consent or is withdrawn from the study and does not complete the follow-up phone call, all subjects must be followed until EOS. Subjects with AEs that are assessed as related to study drug by the Investigator (or designee) which are ongoing at EOS may continue to be followed until the symptoms or value(s) return to normal, or acceptable levels, as judged by the Investigator (or designee) and confirmed by the Sponsor. The Investigator (or designee) should use appropriate judgment in ordering additional tests as necessary to monitor the resolution of events. The Sponsor may request that additional safety tests be performed.

Subjects will receive a follow-up phone call 7 days ( $\pm$  2 days) after EOT or ET to determine if any SAE or drug-related AE has occurred since the EOT or ET visit.

At all times, a subject may be required to remain at the CRU for longer at the discretion of the Investigator (or designee).

Any event that meets the criteria of a suspected unexpected serious adverse reaction will be reported to the institutional review board (IRB) according to CRU policy by the Investigator (or designee) and to regulatory authorities by the Sponsor (or Sponsor designee) according to regulatory authority requirements. Refer to Reference Safety Information in the current IB<sup>1</sup> for pirtobrutinib for additional safety information.

## 7.2.2. Clinical Laboratory Evaluations

Clinical laboratory evaluations (clinical chemistry panel [fasted at least 8 hours; at ET or the day before EOT, subjects are not required to be fasted prior to clinical laboratory evaluations], coagulation parameters, hematology panel, TSH [Screening only], HbA1c [Screening only], CrCl [Screening and Check-in (Day -1)], and UA) will be collected at the timepoints specified in Appendix 4.

Screens for HCV antibody, HBsAg, HBV IgM core antibody, and HIV antibody will be performed at Screening.

Testing for COVID-19 via PCR (or equivalent) will be performed at the timepoints specified in Appendix 4. Testing for COVID-19 may also be conducted periodically during the subject's CRU confinement, at the discretion of the Investigator (or designee). Further details regarding COVID-19 testing (including procedures for subjects who test positive at any time throughout CRU confinement) are specified in a separate document.

A urine drug screen for selected drugs of abuse (including cotinine) and an alcohol screen (urine or breath) will be performed at Screening and repeated at Check-in (Day -1) for all subjects. A serum qualitative or urine qualitative pregnancy test (female subjects only [quantitative serum human chorionic gonadotropin tests may be used for confirmation as needed and post-menopausal subjects may be eligible for participation if the results of the qualitative serum pregnancy or qualitative urine pregnancy test are positive but the quantitative serum human chorionic gonadotropin results are within the laboratory's

reference ranges for post-menopausal women]) and an FSH test (post-menopausal female subjects only) will be performed at the timepoints specified in Appendix 4.

The number of blood samples and total blood volume required for clinical laboratory evaluations are presented in Appendix 3. A list of the specific evaluations is in Appendix 2.

### 7.2.3. Vital Signs

Vital sign measurements (including body temperature, respiratory rate, oxygen saturation, and supine BP and pulse rate) will be obtained at the timepoints specified in Appendix 4.

Blood pressure and pulse rate measurements should be performed using the same arm for each reading and measurements should be taken after the subject has been resting in the supine position for at least 5 minutes.

When vital sign measurements are scheduled at the same time as PK blood draws, the PK blood draws will be obtained at the scheduled timepoint, and the vital sign measurements will be obtained prior to and as close as possible to the scheduled PK blood draw.

## 7.2.4. 12-lead Electrocardiogram

A 12-lead ECG (including HR, PR, RR, QRS, and QT interval parameters) will be obtained after the subject has been resting for at least 10 minutes in the supine position at the timepoints specified in Appendix 4. The QT interval will be corrected for HR by Fridericia's  $(QTcF = QT/[RR]^{1/3})$  formula.

When 12-lead ECGs are scheduled at the same time as PK blood draws, the PK blood draws will be obtained at the scheduled timepoint, and the 12-lead ECGs will be obtained prior to and as close as possible to the scheduled PK blood draw.

### 7.2.5. Physical Examination

A complete or abbreviated physical examination will be performed at the timepoints specified in Appendix 4. Complete physical examinations will evaluate general appearance and the following body systems/organs: dermatological; head and eyes; ears, nose, mouth, and throat; pulmonary; cardiovascular; abdominal; lymphatic; musculoskeletal/extremities; and neurological. Weight and height will be reported (height only reported during Screening). Abbreviated physical examinations will evaluate general appearance and the following body systems/organs: dermatological; pulmonary; cardiovascular; abdominal; and neurological.

## 8. SAMPLE SIZE AND DATA ANALYSIS

#### 8.1. Determination of Sample Size

Up to 28 healthy adult male and female subjects (women of non-childbearing potential only) will be enrolled. This is a relative bioavailability study; however, a total of 28 evaluable subjects (14 subjects per treatment sequence) will provide at least 81% power to have the respective 90% confidence intervals (CIs) for the geometric mean ratios for C<sub>max</sub> and AUC values between test and reference lot tablets are within the interval of 80.00% to 125.00%,

assuming a within subject coefficient of variation (CV) of 25% and that the expected ratio of means is 1.05 (or 0.95). Based on PK results of LOXO-BTK-20009, CV% of AUC is around 25%. Replacement subjects may be enrolled only if deemed necessary by the Sponsor. Every attempt will be made to enroll at least 3 subjects of each sex in the study.

## 8.2. Analysis Populations

## 8.2.1. Pharmacokinetic Population

The PK population will include all subjects who have received a dose of study drug, have at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter can be computed. A subject may be excluded from the PK summary statistics and statistical analysis if the subject has an AE of vomiting that occurs on or before t<sub>max</sub>. The impact of protocol deviations on the PK population will be evaluated on a case-by-case basis.

### 8.2.2. Safety Population

The safety population will consist of all subjects who have received at least 1 dose of study drug. Subjects will be classified into groups based on actual treatment received.

## 8.3. Pharmacokinetic Analysis

Serial PK blood samples for the analysis of plasma concentrations of pirtobrutinib and for future potential and/or exploratory analysis will be collected from predose through 168 hours postdose for each treatment. Whenever possible, the following PK parameters will be calculated for each subject, based on the plasma concentrations of pirtobrutinib (as appropriate):

- AUC<sub>0-24</sub>
- AUC<sub>0-t</sub>
- AUC<sub>0-inf</sub>
- %AUC<sub>extrap</sub>
- CL/F
- t<sub>1/2</sub>
- C<sub>max</sub>
- t<sub>max</sub>
- $\bullet$   $\lambda_z$
- $V_z/F$ .

Pharmacokinetic calculations will be performed using commercial software such as Phoenix<sup>™</sup> WinNonlin<sup>®</sup> Version 8.1 or higher (Certara USA Inc.).

Other parameters may be added as appropriate. Final PK parameters reported will be detailed in the statistical analysis plan (SAP).

Pharmacokinetic analysis will use actual times as recorded on the eCRF. All statistical analyses will be performed using SAS® Version 9.4 or greater. More details on the analyses will be included in the SAP.

### 8.3.1. Descriptive Analysis

Plasma concentrations and PK parameters will be summarized with descriptive statistics (number, arithmetic mean, standard deviation, CV%, geometric mean, geometric CV%, median, minimum, and maximum) by treatment.

Individual and mean plasma concentration-time curves (both linear and log linear) will be included in the final report.

### 8.3.2. Statistical Methodology

The primary PK analysis planned for this study is a mixed effect model including planned treatment sequence, period, and actual treatment as fixed effects and subject within planned treatment sequence as a random effect will be used to analyze the natural log-transformed PK parameters (AUC<sub>0-t</sub>, AUC<sub>0-inf</sub>, and C<sub>max</sub>) and will include calculation of least squared (LS) means and the difference between treatment LS means, as well as their corresponding 90% CIs. The geometric mean ratios and their 90% CIs of the PK parameter for each treatment comparison will be constructed using the exponentiation of the difference and the CIs from the mixed effect model. The comparison of interest is Treatment T (as test) compared with Treatment R (as reference).

#### 8.4. Safety Analysis

All safety assessments, including AEs, SAEs, vital sign measurements, clinical laboratory results, physical examination results, concomitant medications, and 12-lead ECGs, will be tabulated and summarized where possible, using descriptive methodology, as needed, by timepoint. Unless otherwise specified, baseline value is defined as the last non-missing measurement before administration of study drug for each period (ie, Day 1 and Day 8). No formal statistical analyses are planned for the safety data. All safety data will be listed by subject.

Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary (WHO Drug Global B3, September 2019). Adverse events will be coded using Medical Dictionary for Regulatory Activities Version 22.1 (or higher). The incidence of AEs will be presented by severity and by relationship to study drug as determined by the Investigator or designee (Appendix 1 for AE reporting). All TEAEs will be summarized by system organ class and preferred term.

### 8.5. Data Handling and Record Keeping

Any changes to information in the trial progress notes and other source documents will be initialed and dated on the day the change is made by a CRU staff member authorized to make the change. Changes will be made by striking a single line through erroneous data and clearly entering the correct data (eg, wrong data right data). If the reason for the change is not

apparent, a brief explanation for the change will be written adjacent to the change by the CRU staff member.

The Data Management Plan will be approved by the Sponsor.

Data will be validated during data entry by the CRU and verified by the Study Monitor. Data will then be reviewed by the data management group to resolve any outstanding issues. Listings will be generated after the database is cleaned by data management and will be reviewed by the Labcorp Drug Development scientific team. The eCRF and ancillary data will be converted into final SAS® datasets following Study Data Tabulation Model or Sponsor-provided specifications. The final datasets structure will be verified using Web Submission Data Manager®, while the dataset content will be peer reviewed by an independent programmer.

The tables, figures, and listings (TFLs) will be programmed per the final SAP. All TFLs will be peer reviewed by an independent programmer. In addition, draft TFLs will be reviewed by the Labcorp Drug Development scientific team during the dry run and data review meetings.

The peer review will be performed by independent programmers following the quality control process and programming checklists.

## **8.6.** Quality Control and Quality Assurance

Quality control and quality assurance will be performed according to Labcorp Drug Development SOPs or per Sponsor request, and as applicable, according to the contract between Labcorp Drug Development and the Sponsor.

#### 9. ADMINISTRATIVE ASPECTS

### 9.1. Change in Protocol

There will be no alterations in the protocol without agreement between the Sponsor and the Investigator (or designee).

There will be no alterations in the protocol affecting subject safety without the express written approval of the Sponsor, Investigator (or designee), and the IRB (see Form FDA 1572).

### 9.2. Site Initiation Visit/Investigator Meeting

Prior to the start of the clinical study, the representative(s) of the Sponsor and/or Sponsor will meet with the Investigator (or designee) and appropriate CRU staff to familiarize the Investigator (or designee) and CRU staff with the materials necessary for conducting the clinical study.

#### 9.3. Disclosure

All information provided regarding the study, as well as all information collected/documented during the study, will be regarded as confidential. The Investigator (or designee) agrees not to disclose such information in any way without prior written permission from the Sponsor.

Any publication of the results, in part or in total (eg, articles in journals or newspapers, oral presentations, abstracts) by the Investigator (or designee) or their representative(s), shall require prior notification and review, within a reasonable timeframe, by the Sponsor, and cannot be made in violation of the Sponsor's confidentiality restrictions or to the detriment of the Sponsor's intellectual property rights.

### 9.4. Monitoring

The Sponsor will designate a Study Monitor(s) who will be responsible for monitoring this clinical trial. The Sponsor's Study Monitor(s) will monitor the study conduct, proper eCRF and source documentation completion and retention, and accurate study drug accountability. To this end, the Sponsor's Study Monitor(s) will visit the CRU(s) at suitable intervals (or may perform activities remotely as per the Monitoring Plan for this study) and be in frequent contact with the Investigator (or designee) and the Investigator's staff through verbal and written communication. It is essential that the Sponsor's Study Monitor(s) has access to all documents (related to the study and the individual participants) at any time these are requested. In turn, the Sponsor's Study Monitor(s) will adhere to all requirements for subject confidentiality as outlined in the ICF. The Investigator (or designee) and Investigator's staff will be expected to cooperate with the Sponsor's Study Monitor(s), to be available during a portion of the monitoring visit to answer questions, and to provide any missing information.

#### 9.5. Institutional Review Board

In accordance with US Title 21 Code of Federal Regulations (CFR) 56, the protocol, advertisement, ICF, and other information provided to subjects will be reviewed and approved by the IRB. The Sponsor will supply relevant material for the Investigator (or designee) to submit to the IRB for the protocol's review and approval. Verification of the IRB unconditional approval of the protocol and the written ICF statement will be transmitted to the Investigator (or designee).

The IRB will be informed by the Investigator (or designee) of subsequent protocol amendments and of serious and unexpected AEs. Approval for protocol amendments will be transmitted in writing to the Investigator (or designee). If requested, the Investigator (or designee) will permit audits by the IRB and regulatory inspections by providing direct access to source data/documents.

The Investigator (or designee) will provide the IRB with progress reports at appropriate intervals (not to exceed 1 year) and a Study Progress Report following the completion, termination, or discontinuation of the Investigator's (or designee's) participation in the study.

### 9.6. Informed Consent

Written informed consent for the study will be obtained from all subjects before protocol-specific procedures are carried out. The ICF will be approved (along with the protocol) by the IRB and will be acceptable to the Sponsor.

The Investigator (or designee) will explain the nature of the study and the action of the test product. The subjects will be informed that participation is voluntary and that they can withdraw from the study at any time. In accordance with 21 CFR 50, the informed consent process shall be documented by the use of a written ICF approved by the IRB and signed by the subject prior to protocol-specific procedures being performed.

The subject will sign 2 copies of the ICF. One copy will be given to the subject, and the other will be maintained with the subject's records.

#### 9.7. Records

The results from data collected at Screening and during the study will be recorded in the subject's eCRF. To maintain confidentiality, the subjects will be identified only by numbers.

The completed eCRFs will be transferred to the Sponsor (or designee). Copies of each eCRF will be retained by the Investigator (or designee). All source documents, records, and reports will be retained by the CRU in accordance with 21 CFR 312.62(c).

All primary data, or copies thereof (eg, laboratory records, eCRFs, data sheets, correspondence, photographs, and computer records), which are a result of the original observations and activities of the study and are necessary for the reconstruction and evaluation of any study report, will be retained in the CRU archives.

#### 9.8. Reference to Declaration of Helsinki/Basic Principles

The study procedures outlined in this protocol will be conducted in accordance with the US CFR governing Protection of Human Subjects (21 CFR 50), Financial Disclosure by Clinical Investigators (21 CFR 54), IRBs (21 CFR 56), and Investigational New Drug Application (21 CFR 312), as appropriate. As such, these sections of US Title 21 CFR, along with the applicable International Council for Harmonisation Guidelines, are commonly known as Good Clinical Practices, which are consistent with the Declaration of Helsinki.

## 9.9. Financing and Insurance

Financing and insurance will be addressed in a separate agreement.

### 10. REFERENCES

- 1. Loxo Oncology, Inc. LOXO-305 Investigator's Brochure (Version 4.0). 29 October 2020.
- 2. Brandhuber B, Gomez E, Smith S, Eary T, Spencer S, Rothenberg SM, et al. A next generation reversible BTK Inhibitor, for overcoming acquired resistance to irreversible BTK inhibitors. Clin Lymphoma Myeloma Leuk. 2018;18; S216.
- 3. Byrd JC, Furman RR, Coutre SE, Flinn IW, Burger JA, Blum KA, et al. Targeting BTK with ibrutinib in relapsed chronic lymphocytic leukemia. N Engl J Med. 2013 Jul 4;369(1):32–42.
- 4. Woyach JA, Ruppert AS, Guinn D, Lehman A, Blachly JS, Lozanski A, et al. BTKC481S-Mediated Resistance to Ibrutinib in Chronic Lymphocytic Leukemia. J Clin Oncol Off J Am Soc Clin Oncol. 2017 May 1;35(13):1437–43.
- 5. Woyach J, Huang Y, Rogers K, Bhat SA, Grever MR, Lozanski A, et al. Resistance to acalabrutinib in CLL is mediated primarily by BTK mutations. Blood. 2019;134(Supplement 1).
- 6. Chiron D, Di Liberto M, Martin P, Huang X, Sharman J, Blecua P, et al. Cell-cycle reprogramming for PI3K inhibition overrides a relapse-specific C481S BTK mutation revealed by longitudinal functional genomics in mantle cell lymphoma. Cancer Discov. 2014 Sep;4(9):1022–35.
- 7. Xu L, Tsakmaklis N, Yang G, Chen JG, Liu X, Demos M, et al. Acquired mutations associated with ibrutinib resistance in Waldenström macroglobulinemia. Blood. 2017 04;129(18):2519–25.
- 8. Toyoshima S, Kanno A, Kitayama T, Sekiya K, Nakai K, Haruna M, et al. QT PRODACT: In Vivo QT Assay in the Conscious Dog for Assessing the Potential for QT Interval Prolongation by Human Pharmaceuticals [Internet]. Journal of pharmacological sciences. 2005 [cited 2020 Jun 10]. Available from: https://pubmed.ncbi.nlm.nih.gov/16493187/

Protocol CONFIDENTIAL Labcorp Drug Development Study: 8478595 Protocol Reference: LOXO-BTK-21050

# 11. APPENDICES

### **Appendix 1: Adverse Event Reporting**

#### **Adverse Events**

### Definition of Adverse Events

An adverse event (AE; or adverse experience) is defined as any untoward medical occurrence experienced by a patient or healthy adult subject, whether or not considered drug-related by the Investigator (or designee). A treatment-emergent AE is an AE that starts on or after the first administration of study drug.

The following are all AEs:

- unfavorable changes in general condition
- subjective or objective signs/symptoms
- concomitant diseases or accidents
- clinically significant adverse changes in laboratory parameters observed in a subject during a clinical study.

Adverse events comprise all disturbances of general health status, subjective and objective disease symptoms (including laboratory abnormalities that are deemed clinically significant by the Investigator [or designee]), and accidents observed in the context of a clinical trial, irrespective of a possible causal relationship with the administration of the trial substance.

### Categorization of Adverse Events

The severity of AEs will be categorized based on the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 as follows:

- **Grade 1 Mild:** Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
- **Grade 2 Moderate:** Minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL)\*
- Grade 3 Severe or medically significant but not immediately life-threatening: Hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL\*\*
- **Grade 4 Life-threatening consequences:** An event that puts the subject at immediate risk of death
- **Grade 5:** Death related to AE

Note: Not all grades are appropriate for all AEs. Therefore, some AEs are listed within the CTCAE with fewer than 5 options for grade selection. Grade 5 (death) is not appropriate for some AEs and therefore is not an option.

<sup>\*</sup> Instrumental ADL refer to preparing meals, shopping for groceries, or clothes, using the telephone, managing money, etc.

<sup>\*\*</sup>Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

The Investigator (or designee) will make a determination of the relationship of the AE to the study drug using a 2-category system according to the following guidelines:

- **NOT RELATED** = The time course between the administration of investigational product and the occurrence or worsening of the AE rules out a causal relationship and another cause (eg, concomitant drugs, therapies, complications, comorbidities) is suspected.
- **RELATED** = The time course between administration of investigational product and the occurrence or worsening of the AE is consistent with a causal relationship and no other cause (eg, concomitant drugs, therapies, complications, comorbidities) can be identified.

An AE is associated with the use of the drug if there is a reasonable possibility that the experience may have been caused by the drug.

#### Pregnancy

As information is available, a pregnancy (including pregnancy in female partners of male subjects) diagnosed through End of Study or Early Termination (ET; if the subject discontinues from the study and does not complete a follow-up phone call) and for up to 90 days after study drug administration on Day 8 (or last administration of study drug if subject terminates from the study early) should be reported by the Investigator (or designee) via email to Labcorp Drug Development or the Sponsor's Clinical Safety Representative within 24 hours of being notified. Labcorp Drug Development or the Sponsor's Clinical Safety Representative will then forward the Pregnancy Form to the Investigator (or designee) for completion.

## email: SAEIntake@labcorp.com

A subject becoming pregnant while on study drug will immediately be withdrawn from the study and ET study procedures will be performed. The subject or partner should be followed by the Investigator (or designee) until completion of the pregnancy. If the pregnancy ends for any reason before the anticipated date, the Investigator (or designee) should notify Labcorp Drug Development or the Sponsor's Clinical Safety Representative. At the completion of the pregnancy, the Investigator (or designee) will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for immediate classification as a serious adverse event (SAE; ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), the Investigator (or designee) should follow the procedures for reporting an SAE.

Male subjects will be instructed to notify the Investigator (or designee) immediately if they discover their sexual partner is pregnant. In this instance, the partner must provide written consent before pregnancy information can be collected. When a Clinical Research Unit (CRU) becomes aware that the female partner of a male subject is pregnant, they are to contact the Investigator (or designee) immediately (within 24 hours of the CRU staff becoming aware of the event) in addition to notifying Labcorp Drug Development or the Sponsor's Clinical Safety Representative via email.

All pregnancies should be recorded on the AE electronic case report form (eCRF; as appropriate), in addition to completion of the required pregnancy forms. If the Investigator (or designee) suspects that a pregnancy was the result of an interaction between the study treatment and the contraceptive method, in addition to the pregnancy the drug interaction should also be captured as a separate AE.

### **Definition of Serious Adverse Events**

An SAE by the Food and Drug Administration (FDA) definition is any adverse drug experience occurring at any dose that results in any of the following outcomes:

- Death
- A life-threatening adverse drug experience (ie, one that places the subject, in the view of the Investigator [or designee], at immediate risk of death)
- Inpatient hospitalization or prolongation of existing hospitalization
- A persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- An important medical event that may require medical or surgical intervention to prevent 1 of the above outcomes.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered SAEs when, based on appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent 1 of the outcomes listed in this definition.

### Unexpected Adverse Drug Reaction

An AE or suspected adverse drug reaction is considered 'unexpected' if the event is not listed in the Reference Safety Information section of the Investigator's Brochure or if it is not listed at the specificity or severity that has been observed for an unapproved investigational medicinal product.

### Reporting

The FDA-reportable AEs are AEs that are associated with the use of the drug and represent events that are assessed as serious, related, and unexpected. The FDA-reportable AEs will be reported by the CRU to the Sponsor and the responsible Institutional Review Board (IRB). Final determination of whether an event represents a suspected unexpected serious adverse reaction (SUSAR) will be the responsibility of the Sponsor.

Within 24 hours of when an AE that is potentially FDA-reportable is first recognized or reported, and within 24 hours of any SAE (regardless of whether the event is assessed as related or unrelated to study drug) being first recognized or reported, Labcorp Drug

Development or the Sponsor's Clinical Safety Representative will be notified by the Investigator (or designee) in writing using the following email address:

### email: SAEIntake@labcorp.com

To report the SAE, the completed report form should be sent by email to Labcorp Drug Development or the Sponsor's Clinical Safety Representative within 24 hours of awareness. Incoming reports are reviewed during normal business hours. Additional reporting instructions and the SAE Report Form are provided in the Study Manual.

The IRB will be notified of any FDA-reportable AE within the timeframe required by the IRB. The IRB Serious and Unexpected Adverse Experience Submission Form will be completed and submitted with the copy of the written confirmation or summary of the AE.

**Appendix 2: Clinical Laboratory Evaluations** 

| appendix 2. Chinear Daboratory Divardations | | |
|---|---|---|
| Clinical Chemistry Panel (Fasted): | Hematology Panel: | Other Tests: |
| Alanine aminotransferase Albumin Alkaline phosphatase Amylase Aspartate aminotransferase Bilirubin (direct and total) Blood urea nitrogen Calcium Chloride Cholesterol Creatine kinase Creatinine Glucose Iron Lipase Magnesium Phosphorus Potassium Sodium Total protein | Hematocrit Hemoglobin Mean corpuscular hemoglobin Mean corpuscular hemoglobin concentration Mean corpuscular volume Platelet count Red blood cell (RBC) count RBC distribution width White blood cell (WBC) count WBC differential (percent and absolute): Basophils Eosinophils Lymphocytes Monocytes Neutrophils | Hemoglobin A1c <sup>b</sup> Thyroid-stimulating hormone <sup>b</sup> Creatinine clearance <sup>a,d</sup> SARs Coronavirus 19 (COVID-19) test Coagulation Parameters: Partial thromboplastin time Prothrombin time International normalized ratio Serology <sup>b</sup> : Hepatitis B surface antigen Hepatitis B virus immunoglobulin M (IgM) core antibody Hepatitis C virus antibody Human immunodeficiency virus antibody |
| Triglycerides Uric acid | | For Female Subjects Only: |
| | Urinalysis: Bilirubin Color and appearance | Pregnancy test (qualitative serum<br>or qualitative urine, quantitative<br>serum human chorionic<br>gonadotropin tests may be used |
| Urine Drug Screen*: Including but not limited to the following: Alcohol (ethanol) <sup>e</sup> Amphetamines Barbiturates Benzodiazepines Cannabinoids Cocaine (metabolite) | Glucose Ketones Leukocyte esterase Nitrite Occult blood pH and specific gravity Protein Urobilinogen Microscopic examination | for confirmation as needed and post-menopausal subjects may be eligible for participation if the results of the qualitative serum pregnancy or qualitative urine pregnancy test are positive but the quantitative serum human chorionic gonadotropin results are within the laboratory's reference ranges for |
| Methadone Opiates Phencyclidine Cotinine | including, but not limited to,<br>bacteria, casts, crystals, epithelial<br>cells, RBCs, and WBCs (if protein,<br>leukocyte esterase, nitrite, or<br>occult blood is positive) | post-menopausal women) <sup>c</sup> Follicle-stimulating hormone (post-menopausal female subjects only) <sup>b</sup> |

- a. Performed at Screening and Check-in (Day -1) only.
- b. Performed at Screening only.
- c. Performed at Screening, Check-in (Day -1), and Day 14 for End of Treatment or Early Termination only.
- d. Calculated using the Cockcroft-Gault equation.
- e. Urine or breath test.

## **Appendix 3: Total Blood Volume**

The following blood volumes will be withdrawn for each subject:

| Assessment | Approximate<br>Blood Volume per<br>Sample (mL) | Maximum Number of<br>Blood Samples | Approximate<br>Total<br>Volume<br>(mL) |
|---|---|---|---|
| Serology | 8.0 | 1 | 8.0 |
| Pirtobrutinib pharmacokinetic sampling and for future potential and/or exploratory analysis | 4.0 | 39 | 156.0 |
| Clinical laboratory evaluations: | | | |
| Hematology <sup>c</sup> | 4.0 | 10 | 110.0 |
| Clinical chemistry <sup>a</sup> | 4.0 | 10 | 110.0 |
| Coagulation | 3.0 | | |
| Serum pregnancy test (female subjects only) <sup>b</sup> | 4.0 | 3 | 12.0 |
| Serum follicle-stimulating hormone (post- menopausal female subjects only) | 4.0 | 1 | 4.0 |
| | | Total: | 290.0 mL |

<sup>&</sup>lt;sup>a</sup> Thyroid-stimulating hormone and creatinine clearance will be assessed as part of the clinical chemistry sample.

If extra blood samples are required, the maximum blood volume to be withdrawn per subject will not exceed 500 mL.

<sup>&</sup>lt;sup>b</sup> Urine pregnancy tests can be used instead of serum pregnancy tests.

<sup>&</sup>lt;sup>c</sup> Hemoglobin A1c will be taken from hematology sample.

**Appendix 4: Schedule of Assessments** 

| | Screening<br>(Days -41 | Check-in<br>(Day -1) | Period 1 | | | | | | | | | P | Clinic<br>Discharge/<br>EOT/ET <sup>s</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Procedures <sup>a</sup> | to -2) | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 7 (± 2)<br>days post<br>EOT/ET <sup>t</sup> |
| Confined to the CRU | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | | | | |
| Medical History | X | X <sup>b</sup> | | | | | | | | | | | | | | | | |
| Height/Weight/BMI | Xc | X | | | | | | | | | | | | | | | | |
| Physical Examination <sup>d</sup> | | X | | | | | | | | | | | | | | | X | |
| 12-lead ECG <sup>e</sup> | X | X | X | | | | | | | X | | | | | | | X | |
| Vital Sign Measurements <sup>f,g</sup> | X | X | X | | | X | | | | X | | | X | | | | X | |
| HDYF? Inquiry <sup>h</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| AEs/SAEs <sup>i</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pirtobrutinib Dosing | | | $X^{j}$ | | | | | | | $X^k$ | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | | | |
| Clinical Laboratory Evaluations <sup>m</sup> | X | X | | | | X | | | X | | | | X | | | X | X | |
| Creatinine clearance | X | X | | | | | | | | | | | | | | | | |
| Hepatitis and HIV Screen | X | | | | | | | | | | | | | | | | | |
| COVID-19 Screen <sup>n</sup> | X | X | | | | | | | | | | | | | | | | |
| HbA1c Test | X | | | | | | | | | | | | | | | | | |
| Drug Screen <sup>o</sup> | X | X | | | | | | | | | | | | | | | | |
| Prior and Concomitant Medications <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Test <sup>q</sup> | X | X | | | | | | | | | | | | | | X | X | |
| FSH Test <sup>r</sup> | X | | | | | | | | | | | | | | | | | |
| TSH Test | X | | | | | | | | | | | | | | | | | |

Abbreviations: AE = adverse event; BMI = body mass index; COVID-19 = SARS-CoV-2; CRU = Clinical Research Unit; ECG = electrocardiogram; EOS = End of Study; EOT = End of Treatment; ET = Early Termination; FSH = follicle-stimulating hormone; HbA1c = hemoglobin A1c; HDYF? = How Do You Feel?; HIV = human immunodeficiency virus; ICF = Informed Consent Form; PK = pharmacokinetic; SAE = serious adverse event; TSH = thyroid-stimulating hormone; UA = urinalysis.

- a. For details on study procedures, see Section 7.
- b. Interim medical history only.
- c. Height and BMI collected at Screening only.
- d. A complete physical examination will be performed at Check-in (Day -1). An abbreviated physical examination will be performed at Day 15 (EOT) or at ET.
- e. 12-lead ECGs will be obtained at Screening and Check-in (Day -1), Day 1 (predose, and 2 and 4 hours postdose), Day 8 (predose, and 2 and 4 hours postdose), and Day 15 (168 hours postdose on Day 8 [EOT]) or ET. 12-lead ECGs will be collected after the subject has rested in the supine position for at least 10 minutes. When scheduled at the same time as PK blood draws, 12-lead ECGs will be obtained prior to and as close as possible to having blood drawn. The allowed sampling window for 12-lead ECGs is ± 30 minutes from the nominal timepoint for all postdose 12-lead ECGs and no less than 10 minutes prior to dosing for predose 12-lead ECGs.
- f. Vital sign measurements (supine blood pressure and pulse rate) will be obtained at Screening, Check-in (Day -1), Day 1 (predose, and 2 and 4 hours postdose), Day 4 (72 hours postdose on Day 1), Day 8 (predose, and 2 and 4 hours postdose), Day 11 (72 hours on Day 8), and Day 15 (168 hours postdose on Day 8 [EOT]) or ET. Blood pressure and pulse rate will be measured using the same arm for each reading after the subject has been supine for at least 5 minutes. When scheduled at the same time as PK blood draws, vital sign measurements should be carried out prior to and as close as possible to having blood drawn. The allowed sampling window for vital sign measurements is ± 30 minutes from the nominal timepoint for all postdose vital sign measurements and no less than 10 minutes prior to dosing for predose vital sign measurements.
- g. Respiratory rate, oxygen saturation, and body temperature will be obtained at Screening, Check-in (Day -1), and Day 15 (168 hours postdose on Day 8 [EOT]) or ET. Oxygen saturation will also be obtained at predose on Day 1. The allowed sampling window for oxygen saturation measurements is ± 30 minutes from the nominal timepoint for all postdose oxygen saturation measurements and no less than 10 minutes prior to dosing for predose oxygen saturation measurements.
- h. A HDYF? inquiry will be performed at Screening (after the ICF is signed), at Check-in (Day -1), at each postdose vital sign measurement, and at an appropriate time for all other days.
- i. Adverse events and SAEs will be collected beginning at informed consent. Adverse events will be recorded throughout the study (ie, from signing of the ICF until EOS, or until ET if the subject discontinues from the study and does not complete a follow-up phone call), either as subject medical history (if the event is reported as beginning prior to signing of the ICF or if the event occurs prior to study drug administration on Day 1 and is assessed as not related to study procedures by the Investigator [or designee]) or as AEs (if the event occurs after signing of the ICF but prior to study drug administration on Day 1 and is assessed by the Investigator [or designee]) as related to study procedures, or if the event occurs after study drug administration on Day 1 through EOT or ET regardless of relationship to study drug). From EOT or ET through EOS, only AEs assessed as related to study drug are to be recorded. All SAEs that develop from the time of ICF signing until EOS (or ET if the subject discontinues from the study and does not complete a follow-up phone call) are to be reported.
- j. On Day 1, pirtobrutinib will be administered in the morning, either as 2 × 100 mg test lot tablets (total dose 200 mg) or 2 × 100 mg (total dose 200 mg) reference lot tablets following a fast of at least 10 hours predose and 4 hours postdose (with water restricted for 1 hour prior to and 1 hour post-pirtobrutinib administration), according to the treatment sequence the subject is randomly assigned to.
- k. On Day 8, pirtobrutinib will be administered in the morning at approximately the same time as pirtobrutinib was administered on Day 1 (± 15 minutes), either as 2 × 100 mg test lot tablets (total dose 200 mg) or 2 × 100 mg (total dose 200 mg) reference lot tablets following a fast of at least 10 hours predose and 4 hours postdose (with water restricted for 1 hour prior to and 1 hour post-pirtobrutinib administration), according to the treatment sequence the subject is randomly assigned to.

CCI

m. Clinical chemistry panel (fasted for at least 8 hours), coagulation parameters, hematology panel, and UA will be performed at Screening, Check-in (Day -1), Day 4 (72 hours postdose on Day 1), Day 7 (144 hours postdose on Day 1), Day 11 (72 hours postdose on Day 8), and Day 14 (144 hours postdose on Day 8, if the subject completes the study [EOT]), or on the day of ET. At ET or the day before EOT (Day 14), subjects are not required to be fasted prior to clinical laboratory evaluations.

- CONFIDENTIAL Protocol Reference: LOXO-BTK-21050
- n. Testing for COVID-19 will be conducted at a minimum at Screening and Check-in (Day -1). Testing for COVID-19 may also be conducted periodically during the subject's CRU
- o. Urine drug screen for selected drugs of abuse (including cotinine) and alcohol screen (urine or breath).
- p. Prior and concomitant medication administration will be recorded beginning at informed consent. In addition, all Investigator-approved prescription and over-the-counter medications taken by a subject within 14 days or 5 half-lives (if known), whichever is longer, prior to Day 1 will be recorded on the subject's electronic case report form.
- q. Female subjects only. Performed at Screening, Check-in (Day -1), and Day 14 (144 hours postdose on Day 8), if the subject completes the study (EOT) or on the day of ET.

confinement, at the discretion of the Investigator (or designee). Tests will be performed by rapid polymerase chain reaction or equivalent.

- r. Post-menopausal female subjects only.
- s. End of Treatment is defined as when the subject is released from the CRU following completion of all assessments through Day 15. Early Termination is defined as when the subject is released from the CRU if the subject terminates the study early. Vital sign measurements, ECG, and abbreviated physical examination results are to be available for review by the Investigator (or designee) prior to subject release from the CRU on Day 15 (EOT) or ET. Clinical laboratory results (for clinical chemistry, hematology, coagulation, and UA) and pregnancy test results (female subjects only) are to be available for review by the Investigator (or designee) prior to subject release from the CRU at the ET visit, if available.
- t. To be conducted 7 days (± 2 days) following EOT or ET. End of Study is defined as when the subject is contacted by the CRU for a follow-up phone call 7 days (± 2 days) after the EOT visit or ET visit to determine if any SAE or study drug-related AE has occurred since the EOT or ET visit. All subjects who received pirtobrutinib (including subjects who are terminated early) will receive a follow-up phone call.